CLINICAL TRIAL: NCT04546425
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE GIVEN AS A SERIES OF 2 INFANT DOSES AND 1 TODDLER DOSE IN HEALTHY INFANTS
Brief Title: 20-valent Pneumococcal Conjugate Vaccine Safety and Immunogenicity Study of a 3-Dose Series in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B7471012; 2019-003306-27 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-09-14 (Actual); Results first posted 2023-05-15 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20-valent pneumococcal conjugate vaccine (Experimental): Pneumococcal conjugate vaccine
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine
- 13-valent pneumococcal conjugate vaccine (Active Comparator): Pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine — 20-valent pneumococcal conjugate vaccine
  Arms: 20-valent pneumococcal conjugate vaccine
Biological: 13-valent pneumococcal conjugate vaccine — 13-valent pneumococcal conjugate vaccine
  Arms: 13-valent pneumococcal conjugate vaccine

SUMMARY:
20-valent Pneumococcal Conjugate Vaccine Safety and Immunogenicity Study of a 3-Dose Series in Healthy Infants

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants born at >36 weeks of gestation and 2 months of age at the time of consent.
* Healthy infants determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis).
* Major known congenital malformation or serious chronic disorder.
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.

Ages: 42 Days to 112 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1258 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2023-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (66):
- Australia (2):
  - Perth Children's Hospital, Nedlands, Western Australia
  - Telethon Kids Institute, Vaccine Trials Group, Perth Children's Hospital, Nedlands, Western Australia
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Antwerp, Edegem
- Czechia (7):
  - DD ordinace s.r.o., Jindřichův Hradec
  - Ordinace praktického lékaře pro děti a dorost, Jindřichův Hradec
  - Samostatna ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Zdravotnicke stredisko Dubina, verejna obchodni spolecnost, Pardubice
  - MUDr. Jitka Fabianova, Prague
  - MEDICENTRUM 6 s.r.o. - Ordinace praktickeho lekare pro deti a dorost, Prague
  - Medicentrum 6 s.r.o., Prague
- Hvidovre Hospital, Hvidovre, Denmark
- Estonia (6):
  - Kadrina Tervisekeskus OU, Kadrina
  - Merekivi Perearstid., Tallinn
  - Merelahe Family Doctors Centre, Tallinn
  - OU Al Mare Perearstikeskus, Tallinn
  - Sinu Arst Health Center, Tallinn
  - Clinical Research Centre, Tartu
- Finland (11):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Jarvenpaa Vaccine Research Clinic, Jarvenpaa
  - Kokkola Vaccine Research Clinic, Kokkola
  - FVR, Oulun rokotetutkimusklinikka, Oulu
  - Tampereen yliopisto Oulun Rokotetutkimusklinikka, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinäjoki Vaccine Research Clinic, Seinäjoki
  - Tampere Vaccine Research Center, Tampere
  - Turku Vaccine Research Clinic, Turku
- Italy (4):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico U.O.S.D. Pediatria Alta lntensita di Cura, Milan, Milan
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - Azienda Ospedaliera Universitaria, Foggia
  - Ospedale Policlinico San Martino, Genova
- Netherlands (2):
  - Stichting Apotheek der Haarlemse Ziekenhuizen, Haarlem
  - Spaarne Gasthuis (Kennemer Gasthuis), Hoofddorp
- Norway (4):
  - Akershus University Hospital, Lorenskog
  - Oslo University Hospital, Ulleval, Oslo
  - Stavanger University Hospital, Stavanger
  - Akershus University Hospital - Sykehusapoteket Ahus, Viken
- Poland (16):
  - IN-VIVO Sp z o.o. IN-VIVO Bydgoszcz, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Prywatny Gabinet Lekarski dr n. med. Jerzy Brzostek, Dębica
  - Centrum Badan Klinicznych JCI, Krakow
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II Oddzial Pediatrii i Neurologii Dzieciecej, Krakow
  - GRAVITA. Diagnostyka i Leczenie nieplodnosci, Lodz
  - Rodzinne Centrum Medyczne LUBMED, Luboń
  - Specjalistyczny Zespół Opieki Zdrowotnej nad Matką i Dzieckiem w Poznaniu, Poznan
  - Niepubliczny Zaklad Lecznictwa Ambulatoryjnego Michalkowice Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie
  - Nasz Lekarz Przychodnie Medyczne Slawomir Jeka, Torun
  - Szpital im. Sw. Jadwigi Slaskiej w Trzebnicy, Trzebnica
  - Szpital Bielanski im. ks. J. Popieluszki SPZOZ, Warsaw
  - Provita 001, Warsaw
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego we Wroclawiu, Wroclaw
  - Centrum Medyczne AD-MED Sp. z o. o. Przychodnia Dla Rodziny, Wroclaw
  - Niepubliczny Zaklad Opieki Zdrowotnej "SALMED", Łęczna
- Russia (4):
  - Federal State Budget Institution of Healthcare Central clinical hospital of Russian, Moscow
  - State Budget Institution of Healthcare of Perm Region "City Children's Clinical Polyclinic #5", Perm
  - LLC PiterClinica, Saint Petersburg
  - State autonomous institution of healthcare of Sverdlovsk region, Yekaterinburg
- Slovakia (7):
  - PEDIAMED s.r.o., Bratislava
  - NASA DOKTORKA s.r.o., Bratislava
  - Rozvojova agentura Banskobystrickeho samospravneho kraja, n.o., Detva
  - MUDr. Martin Zavrel Vseobecna ambulancia pre deti a dorast, Horné Srnie
  - Všeobecná ambulancia pre deti a dorast, Humenné
  - PEDAMB s.r.o., Košice
  - MUDr. Drusková s.r.o., Liptovská Osada

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Senders S, Korbal P, Kline M, Tamimi N, Thompson A, Drozd J, Cutler MW, Giardina PC, Trammel J, Lei L, Peng Y, Watson W, McElwee K. Immunogenicity and safety of concomitant vaccines given with 20-valent pneumococcal conjugate vaccine in healthy infants. Vaccine. 2025 Dec 5;68:127916. doi: 10.1016/j.vaccine.2025.127916. Epub 2025 Nov 3. PMID 41187484
- [Derived] Korbal P, Wysocki J, Jackowska T, Kline M, Tamimi N, Drozd J, Lei L, Peng Y, Giardina PC, Gruber W, Scott D, Watson W. Phase 3 Safety and Immunogenicity Study of a Three-dose Series of Twenty-valent Pneumococcal Conjugate Vaccine in Healthy Infants and Toddlers. Pediatr Infect Dis J. 2024 Jun 1;43(6):587-595. doi: 10.1097/INF.0000000000004300. Epub 2024 Mar 8. PMID 38456705
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471012

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For primary study population,1207 participants were enrolled and assigned to receive 3 doses of 20-valent pneumococcal conjugate vaccine (20vPnC) or 13-valent pneumococcal conjugate vaccine (13vPnC) of which 3 participants were not vaccinated, 1204 were vaccinated with 20vPnC or 13vPnC.Additional 51 Russian participants were enrolled, all of whom were vaccinated with 20vPnC or 13vPnC.
Groups:
- 20vPnC: Primary Study Population: Infants 42 to 112 days of age were enrolled to receive 3 doses of 0.5 millilitre (mL) 20vPnC intramuscularly. Dose 1 was administered at enrollment, dose 2 was given 42 to 63 days after dose 1 and dose 3 was administered at 11 to 12 months of age.
- 13vPnC: Primary Study Population: Infants 42 to 112 days of age were enrolled to receive 3 doses of 0.5 mL 13vPnC intramuscularly. Dose 1 was administered at enrollment, dose 2 was given 42 to 63 days after dose 1 and dose 3 was administered at 11 to 12 months of age.
- 20vPnC: Russian Cohort: Infants 42 to 70 days of age were enrolled to receive 3 doses of 0.5 mL 20vPnC intramuscularly. Dose 1 was administered at enrollment, dose 2 was given 60 to 90 days after dose 1 and dose 3 was administered at 11 to 15 months of age.
- 13vPnC: Russian Cohort: Infants 42 to 70 days of age were enrolled to receive 3 doses of 0.5 mL 13vPnC intramuscularly. Dose 1 was administered at enrollment, dose 2 was given 60 to 90 days after dose 1 and dose 3 was administered at 11 to 15 months of age.
Period: Overall Study
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Started | 601 | 603 | 24 | 27
Dose 1 | 601 | 603 | 24 | 27
Dose 2 | 593 | 598 | 24 | 27
Dose 3 | 588 | 594 | 22 | 25
Completed | 583 | 590 | 22 | 25
Not Completed | 18 | 13 | 2 | 2
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 4 | 0 | 0
Not completed — No Longer met eligibility criteria | 3 | 3 | 1 | 1
Not completed — Withdrawal by parent/guardian | 6 | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort | Total
Number analyzed (Participants) | 601 | 603 | 24 | 27 | 1255
Age, Customized [Count of Participants; unit: Participants]
  28 days-23 months | 601 | 603 | 24 | 27 | 1255
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 292 | 16 | 12 | 622
  Male | 299 | 311 | 8 | 15 | 633
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 0 | 0 | 5
  Not Hispanic or Latino | 577 | 586 | 22 | 25 | 1210
  Unknown or Not Reported | 20 | 16 | 2 | 2 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 5 | 0 | 1 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 585 | 592 | 24 | 26 | 1227
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 7 | 5 | 0 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 1: Primary Study Population
Description: Local reactions included redness, swelling and, pain at the injection site, recorded by parents/legal guardians of participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild (greater than [>] 0 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7.0 cm). Pain at injection site was graded as mild (hurt if gently touched example, whimpered, winced, protested, or withdrew), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement). 95 percent (%) confidence interval (CI) was based on Clopper and Pearson method.
Time Frame: Within 7 days after Dose 1
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies the number of participants with any e-diary data after Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 598 | 603
Percentage of participants
  Redness: Mild | 20.7 (17.6) [17.6 to 24.2] | 22.7 (19.4) [19.4 to 26.3]
  Redness: Moderate | 4.5 (3.0) [3.0 to 6.5] | 4.8 (3.2) [3.2 to 6.8]
  Redness: Severe | 0 (0.0) [0.0 to 0.6] | 0 (0.0) [0.0 to 0.6]
  Swelling: Mild | 12.7 (10.1) [10.1 to 15.6] | 12.9 (10.4) [10.4 to 15.9]
  Swelling: Moderate | 8.7 (6.6) [6.6 to 11.2] | 7.3 (5.4) [5.4 to 9.7]
  Swelling: Severe | 0 (0.0) [0.0 to 0.6] | 0 (0.0) [0.0 to 0.6]
  Pain at Injection Site: Mild | 16.7 (13.8) [13.8 to 20.0] | 17.9 (14.9) [14.9 to 21.2]
  Pain at Injection Site: Moderate | 12.0 (9.5) [9.5 to 14.9] | 11.4 (9.0) [9.0 to 14.3]
  Pain at Injection Site: Severe | 0.3 (0.0) [0.0 to 1.2] | 0 (0.0) [0.0 to 0.6]

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2: Primary Study Population
Description: Local reactions included redness, swelling and, pain at the injection site, recorded by parents/legal guardians of participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm. Redness and swelling were graded as mild (>0 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7.0 cm). Pain at injection site was graded as mild (hurt if gently touched example, whimpered, winced, protested, or withdrew), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after Dose 2
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies the number of participants with any e-diary data after Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 592 | 594
Percentage of participants
  Redness: Mild | 24.8 (21.4) [21.4 to 28.5] | 22.9 (19.6) [19.6 to 26.5]
  Redness: Moderate | 3.7 (2.3) [2.3 to 5.6] | 5.1 (3.4) [3.4 to 7.1]
  Redness: Severe | 0 (0.0) [0.0 to 0.6] | 0.2 (0.0) [0.0 to 0.9]
  Swelling: Mild | 13.7 (11.0) [11.0 to 16.7] | 14.1 (11.4) [11.4 to 17.2]
  Swelling: Moderate | 8.3 (6.2) [6.2 to 10.8] | 6.2 (4.4) [4.4 to 8.5]
  Swelling: Severe | 0 (0.0) [0.0 to 0.6] | 0.2 (0.0) [0.0 to 0.9]
  Pain at Injection Site: Mild | 13.3 (10.7) [10.7 to 16.4] | 16.5 (13.6) [13.6 to 19.7]
  Pain at Injection Site: Moderate | 9.3 (7.1) [7.1 to 11.9] | 7.9 (5.9) [5.9 to 10.4]
  Pain at Injection Site: Severe | 0.2 (0.0) [0.0 to 0.9] | 0.2 (0.0) [0.0 to 0.9]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3: Primary Study Population
Description: as for outcome 2
Time Frame: Within 7 days after Dose 3
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies the number of participants with any e-diary data after Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 580 | 586
Percentage of participants
  Redness: Mild | 23.3 (19.9) [19.9 to 26.9] | 25.1 (21.6) [21.6 to 28.8]
  Redness: Moderate | 13.4 (10.8) [10.8 to 16.5] | 8.5 (6.4) [6.4 to 11.1]
  Redness: Severe | 0.2 (0.0) [0.0 to 1.0] | 0.2 (0.0) [0.0 to 0.9]
  Swelling: Mild | 17.8 (14.7) [14.7 to 21.1] | 14.5 (11.8) [11.8 to 17.6]
  Swelling: Moderate | 11.9 (9.4) [9.4 to 14.8] | 9.7 (7.5) [7.5 to 12.4]
  Swelling: Severe | 0.2 (0.0) [0.0 to 1.0] | 0.3 (0.0) [0.0 to 1.2]
  Pain at Injection Site: Mild | 24.7 (21.2) [21.2 to 28.4] | 22.4 (19.0) [19.0 to 25.9]
  Pain at Injection Site: Moderate | 17.4 (14.4) [14.4 to 20.8] | 17.2 (14.3) [14.3 to 20.5]
  Pain at Injection Site: Severe | 0.3 (0.0) [0.0 to 1.2] | 0.3 (0.0) [0.0 to 1.2]

4. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1: Primary Study Population
Description: Systemic events: fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participants using an e-diary. Fever: was defined as temperature >=38.0 degree Celsius (C) and categorized as >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0-degree C. Decreased appetite: mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased/prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability: mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 Days after Dose 1
Population: Safety analysis set: all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies number of participants with any e-diary data after Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 598 | 603
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 7.5 (5.5) [5.5 to 9.9] | 6.8 (4.9) [4.9 to 9.1]
  Fever: >38.4 degrees C to 38.9 degrees C | 1.3 (0.6) [0.6 to 2.6] | 1.3 (0.6) [0.6 to 2.6]
  Fever: >38.9 degrees C to 40.0 degrees C | 0 (0.0) [0.0 to 0.6] | 0.3 (0.0) [0.0 to 1.2]
  Fever: >40.0 degrees C | 0 (0.0) [0.0 to 0.6] | 0 (0.0) [0.0 to 0.6]
  Decreased appetite: Mild | 16.2 (13.4) [13.4 to 19.4] | 13.3 (10.7) [10.7 to 16.2]
  Decreased appetite: Moderate | 7.5 (5.5) [5.5 to 9.9] | 8.8 (6.7) [6.7 to 11.3]
  Decreased appetite: Severe | 1.0 (0.4) [0.4 to 2.2] | 0.5 (0.1) [0.1 to 1.4]
  Drowsiness: Mild | 46.0 (41.9) [41.9 to 50.1] | 48.6 (44.5) [44.5 to 52.7]
  Drowsiness: Moderate | 14.4 (11.7) [11.7 to 17.5] | 14.3 (11.6) [11.6 to 17.3]
  Drowsiness: Severe | 0.8 (0.3) [0.3 to 1.9] | 0.8 (0.3) [0.3 to 1.9]
  Irritability: Mild | 17.6 (14.6) [14.6 to 20.8] | 17.4 (14.5) [14.5 to 20.7]
  Irritability: Moderate | 46.2 (42.1) [42.1 to 50.2] | 46.4 (42.4) [42.4 to 50.5]
  Irritability: Severe | 8.2 (6.1) [6.1 to 10.7] | 8.6 (6.5) [6.5 to 11.2]

5. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2: Primary Study Population
Description: Systemic events: fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participant's using an e-diary. Fever: was defined as temperature >=38.0 degree C and categorized as >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0-degree C. Decreased appetite: mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased/prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability: mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 Days after Dose 2
Population: Safety analysis set: all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here," Number of Participants Analyzed" signifies number of participants with any e-diary data after Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 592 | 594
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 11.7 (9.2) [9.2 to 14.5] | 11.6 (9.2) [9.2 to 14.5]
  Fever: >38.4 degrees C to 38.9 degrees C | 2.5 (1.4) [1.4 to 4.1] | 2.0 (1.0) [1.0 to 3.5]
  Fever: >38.9 degrees C to 40.0 degrees C | 0.7 (0.2) [0.2 to 1.7] | 0.3 (0.0) [0.0 to 1.2]
  Fever: >40.0 degrees C | 0 (0.0) [0.0 to 0.6] | 0 (0.0) [0.0 to 0.6]
  Decreased appetite: Mild | 13.5 (10.9) [10.9 to 16.5] | 12.1 (9.6) [9.6 to 15.0]
  Decreased appetite: Moderate | 10.1 (7.8) [7.8 to 12.9] | 6.4 (4.6) [4.6 to 8.7]
  Decreased appetite: Severe | 1.0 (0.4) [0.4 to 2.2] | 0.8 (0.3) [0.3 to 2.0]
  Drowsiness: Mild | 37.8 (33.9) [33.9 to 41.9] | 37.0 (33.1) [33.1 to 41.1]
  Drowsiness: Moderate | 13.2 (10.6) [10.6 to 16.2] | 13.5 (10.8) [10.8 to 16.5]
  Drowsiness: Severe | 0.3 (0.0) [0.0 to 1.2] | 0.2 (0.0) [0.0 to 0.9]
  Irritability: Mild | 22.8 (19.5) [19.5 to 26.4] | 21.2 (18.0) [18.0 to 24.7]
  Irritability: Moderate | 43.1 (39.0) [39.0 to 47.2] | 40.6 (36.6) [36.6 to 44.6]
  Irritability: Severe | 5.7 (4.0) [4.0 to 7.9] | 6.6 (4.7) [4.7 to 8.9]

6. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3: Primary Study Population
Description: Systemic events: fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participants using an e-diary. Fever: was defined as temperature >=38.0 degree C and categorized as >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0-degree C. Decreased appetite: mild (decreased interest in eating), moderate (decreased oral intake) & severe (refusal to feed). Drowsiness was graded as mild (increased/prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability: mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 Days after Dose 3
Population: Safety analysis set: all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here," Number of Participants Analyzed" signifies number of participants with any e-diary data after Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 580 | 586
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 13.4 (10.8) [10.8 to 16.5] | 13.5 (10.8) [10.8 to 16.5]
  Fever: >38.4 degrees C to 38.9 degrees C | 6.9 (5.0) [5.0 to 9.3] | 7.0 (5.1) [5.1 to 9.4]
  Fever: >38.9 degrees C to 40.0 degrees C | 3.6 (2.3) [2.3 to 5.5] | 3.2 (2.0) [2.0 to 5.0]
  Fever: >40.0 degrees C | 0.3 (0.0) [0.0 to 1.2] | 0 (0.0) [0.0 to 0.6]
  Decreased appetite: Mild | 20.0 (16.8) [16.8 to 23.5] | 15.5 (12.7) [12.7 to 18.7]
  Decreased appetite: Moderate | 17.1 (14.1) [14.1 to 20.4] | 18.9 (15.8) [15.8 to 22.4]
  Decreased appetite: Severe | 2.2 (1.2) [1.2 to 3.8] | 2.0 (1.1) [1.1 to 3.5]
  Drowsiness: Mild | 34.8 (30.9) [30.9 to 38.9] | 32.8 (29.0) [29.0 to 36.7]
  Drowsiness: Moderate | 15.3 (12.5) [12.5 to 18.5] | 14.7 (11.9) [11.9 to 17.8]
  Drowsiness: Severe | 0.7 (0.2) [0.2 to 1.8] | 1.2 (0.5) [0.5 to 2.4]
  Irritability: Mild | 23.4 (20.1) [20.1 to 27.1] | 21.3 (18.1) [18.1 to 24.9]
  Irritability: Moderate | 43.4 (39.4) [39.4 to 47.6] | 45.4 (41.3) [41.3 to 49.5]
  Irritability: Severe | 4.1 (2.7) [2.7 to 6.1] | 4.1 (2.6) [2.6 to 6.0]

7. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 1 to 1 Month After Dose 2: Primary Study Population
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. 95% CI was based on the Clopper and Pearson method. AEs reported in this outcome measure excluded local reactions and systemic events collected from an e-diary.
Time Frame: From Dose 1 to 1 month after Dose 2
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 601 | 603
Percentage of participants | 13.8 (11.2) [11.2 to 16.8] | 14.4 (11.7) [11.7 to 17.5]

8. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 3 to 1 Month After Dose 3: Primary Study Population
Description: as for outcome 7
Time Frame: From Dose 3 to 1 month after Dose 3
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies the number of participants who received Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 588 | 594
Percentage of participants | 15.5 (12.6) [12.6 to 18.7] | 16.5 (13.6) [13.6 to 19.7]

9. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Dose 1 to 1 Month After Dose 3: Primary Study Population
Description: A SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; was a congenital anomaly/birth defect and other important medical events. 95% CI was based on the Clopper and Pearson method.
Time Frame: From Dose 1 to 1 month after Dose 3
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 601 | 603
Percentage of participants | 5.7 (3.9) [3.9 to 7.8] | 6.6 (4.8) [4.8 to 8.9]

10. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Condition (NDCMC) From Dose 1 to 1 Month After Dose 3: Primary Study Population
Description: A NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long-lasting in its effects. 95% CI was based on the Clopper and Pearson method.
Time Frame: From Dose 1 to 1 month after Dose 3
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 601 | 603
Percentage of participants | 1.0 (0.4) [0.4 to 2.2] | 1.0 (0.4) [0.4 to 2.2]

11. Primary Outcome: Percentage of Participants With Predefined Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After Dose 2: Primary Study Population
Description: Predefined IgG concentrations were as follows: for serotype 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, 33F: >=0.35 microgram per mL (mcg/mL), for serotype 5: >=0.23 mcg/mL, for serotype 6B: >=0.10 mcg/mL and for serotype 19A: >=0.12 mcg/mL. 95% CI was based on the Clopper and Pearson method.
Time Frame: 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population: eligible participants 42-112 days of age at first vaccination, received first 2 doses as randomized, at least 1 valid immunogenicity results from blood collection (27 to 56 days after Dose 2), no other major protocol deviations. "Number of Participants Analyzed"= participants in Dose 2 evaluable immunogenicity population, "Number Analyzed"= participants with valid IgG assay results for specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 567 | 562
Percentage of participants
  Serotype 1: number analyzed (Participants) | 566 | 562
  Serotype 1 | 70.7 [66.7 to 74.4] | 84.2 [80.9 to 87.1]
  Serotype 3: number analyzed (Participants) | 566 | 562
  Serotype 3 | 58.0 [53.8 to 62.1] | 75.8 [72.0 to 79.3]
  Serotype 4: number analyzed (Participants) | 566 | 562
  Serotype 4 | 68.6 [64.5 to 72.4] | 79.5 [76.0 to 82.8]
  Serotype 5: number analyzed (Participants) | 566 | 562
  Serotype 5 | 63.4 [59.3 to 67.4] | 76.0 [72.2 to 79.5]
  Serotype 6A: number analyzed (Participants) | 566 | 562
  Serotype 6A | 59.5 [55.4 to 63.6] | 73.7 [69.8 to 77.3]
  Serotype 6B: number analyzed (Participants) | 564 | 561
  Serotype 6B | 20.7 [17.5 to 24.3] | 36.5 [32.5 to 40.7]
  Serotype 7F: number analyzed (Participants) | 566 | 562
  Serotype 7F | 87.6 [84.6 to 90.2] | 90.2 [87.5 to 92.5]
  Serotype 9V: number analyzed (Participants) | 566 | 562
  Serotype 9V | 60.2 [56.1 to 64.3] | 74.6 [70.7 to 78.1]
  Serotype 14: number analyzed (Participants) | 565 | 562
  Serotype 14 | 78.6 [75.0 to 81.9] | 81.9 [78.4 to 85.0]
  Serotype 18C: number analyzed (Participants) | 566 | 562
  Serotype 18C | 71.0 [67.1 to 74.7] | 76.5 [72.8 to 80.0]
  Serotype 19A: number analyzed (Participants) | 566 | 562
  Serotype 19A | 92.2 [89.7 to 94.3] | 94.0 [91.6 to 95.8]
  Serotype 19F: number analyzed (Participants) | 566 | 562
  Serotype 19F | 94.3 [92.1 to 96.1] | 95.7 [93.7 to 97.2]
  Serotype 23F: number analyzed (Participants) | 566 | 562
  Serotype 23F | 23.5 [20.1 to 27.2] | 41.8 [37.7 to 46.0]
  Serotype 8: number analyzed (Participants) | 567 | 561
  Serotype 8 | 96.5 [94.6 to 97.8] | 2.9 [1.6 to 4.6]
  Serotype 10A | 28.9 [25.2 to 32.8] | 2.7 [1.5 to 4.4]
  Serotype 11A | 94.2 [91.9 to 96.0] | 2.0 [1.0 to 3.5]
  Serotype 12F | 30.3 [26.6 to 34.3] | 0.2 [0.0 to 1.0]
  Serotype 15B: number analyzed (Participants) | 566 | 562
  Serotype 15B | 94.3 [92.1 to 96.1] | 8.5 [6.4 to 11.2]
  Serotype 22F | 94.4 [92.1 to 96.1] | 2.0 [1.0 to 3.5]
  Serotype 33F: number analyzed (Participants) | 566 | 562
  Serotype 33F | 46.8 [42.6 to 51.0] | 2.7 [1.5 to 4.4]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 1; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC to the corresponding serotype in 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CIs for the percentage differences (20vPnC-13vPnC) was greater than -10%; Percent Difference : = -13.5, 95% CI 2-sided [-18.3 to -8.7] — 2-Sided 95% CIs were calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage
Statistical Analysis 2: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -17.9, 95% CI 2-sided [-23.2 to -12.4] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 3: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -11.0, 95% CI 2-sided [-16.0 to -5.9] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 4: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 5; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -12.6, 95% CI 2-sided [-17.8 to -7.2] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 5: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 6A; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -14.1, 95% CI 2-sided [-19.5 to -8.6] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 6: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -15.8, 95% CI 2-sided [-21.0 to -10.6] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 7: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -2.6, 95% CI 2-sided [-6.3 to 1.1] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 8: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -14.3, 95% CI 2-sided [-19.7 to -8.9] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 9: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 14; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -3.3, 95% CI 2-sided [-7.9 to 1.4] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 10: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -5.5, 95% CI 2-sided [-10.6 to -0.4] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 11: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -1.7, 95% CI 2-sided [-4.8 to 1.3] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 12: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -1.4, 95% CI 2-sided [-4.0 to 1.2] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 13: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 1]; Percent Difference = -18.3, 95% CI 2-sided [-23.6 to -12.9] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 14: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 8; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results are from serotype 6B (13vPnC serotype with the lowest percentage, not including serotype 3) in the 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CIs for the percentage differences (20vPnC - lowest 13vPnC) was greater than -10%; Percent difference = 59.9, 95% CI 2-sided [55.6 to 64.1] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 15: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 10A; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 14]; Percent difference = -7.6, 95% CI 2-sided [-13.1 to -2.1] — 2-Sided 95% CI based on the Percent difference for the difference in proportions expressed as a percentage
Statistical Analysis 16: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 11A; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 14]; Percent difference = 57.6, 95% CI 2-sided [53.1 to 61.9] — 2-Sided 95% CI based on the Percent difference for the difference in proportions expressed as a percentage
Statistical Analysis 17: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 12F; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 14]; Percent difference = -6.2, 95% CI 2-sided [-11.7 to -0.7] — 2-Sided 95% CI based on the Percent difference for the difference in proportions expressed as a percentage
Statistical Analysis 18: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 15B; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 14]; Percent difference = 57.8, 95% CI 2-sided [53.3 to 62.1] — 2-Sided 95% CI based on the Percent difference for the difference in proportions expressed as a percentage
Statistical Analysis 19: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 22F; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 14]; Percent difference = 57.8, 95% CI 2-sided [53.3 to 62.1] — 2-Sided 95% CI based on the Percent difference for the difference in proportions expressed as a percentage
Statistical Analysis 20: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 33F; Test type: Non-Inferiority — [test comment as in outcome 11, analysis 14]; Percent difference = 10.3, 95% CI 2-sided [4.5 to 16.0] — 2-Sided 95% CI based on the Percent difference for the difference in proportions expressed as a percentage

12. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Pneumococcal IgG Antibody 1 Month After Dose 2: Primary Study Population
Description: Pneumococcal serotype-specific IgG concentration was measured for serum sample for 13vPnC serotype: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 7 additional serotype: 8, 10A, 11A, 12F, 15B, 22F, 33F. GMC and corresponding 2-sided 95% CIs were calculated by exponentiating mean logarithm of concentration, corresponding 2-sided 95% CIs (based on Student's t distribution). Assay result below LLOQ was set to 0.5*LLOQ. Geometric mean ratios (GMRs) were reported in statistical analysis section and were calculated by exponentiating mean difference of logarithm of concentration and corresponding 2-sided 95% CIs (based on Student's t distribution).
Time Frame: 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population: eligible participants 42-112 days of age at first vaccination, received 1st 2 doses as randomized, at least 1 valid immunogenicity result from blood collection (27-56 days after Dose2). "Number of Participants Analyzed"=participants in Dose 2 evaluable immunogenicity population, "Number Analyzed"= participants with valid IgG assay result for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per millilitre (mcg/mL)
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 567 | 562
Microgram per millilitre (mcg/mL)
  Serotype 1: number analyzed (Participants) | 566 | 562
  Serotype 1 | 0.57 [0.52 to 0.62] | 0.93 [0.86 to 1.01]
  Serotype 3: number analyzed (Participants) | 566 | 562
  Serotype 3 | 0.41 [0.38 to 0.45] | 0.58 [0.54 to 0.63]
  Serotype 4: number analyzed (Participants) | 566 | 562
  Serotype 4 | 0.55 [0.50 to 0.61] | 0.92 [0.83 to 1.02]
  Serotype 5: number analyzed (Participants) | 566 | 562
  Serotype 5 | 0.34 [0.30 to 0.38] | 0.56 [0.50 to 0.62]
  Serotype 6A: number analyzed (Participants) | 566 | 562
  Serotype 6A | 0.45 [0.40 to 0.52] | 0.84 [0.73 to 0.95]
  Serotype 6B: number analyzed (Participants) | 564 | 561
  Serotype 6B | 0.03 [0.03 to 0.04] | 0.06 [0.05 to 0.07]
  Serotype 7F: number analyzed (Participants) | 566 | 562
  Serotype 7F | 1.02 [0.94 to 1.10] | 1.41 [1.30 to 1.53]
  Serotype 9V: number analyzed (Participants) | 566 | 562
  Serotype 9V | 0.45 [0.40 to 0.51] | 0.77 [0.68 to 0.87]
  Serotype 14: number analyzed (Participants) | 565 | 562
  Serotype 14 | 1.05 [0.94 to 1.18] | 1.28 [1.14 to 1.43]
  Serotype 18C: number analyzed (Participants) | 566 | 562
  Serotype 18C | 0.69 [0.62 to 0.77] | 0.87 [0.78 to 0.98]
  Serotype 19A: number analyzed (Participants) | 566 | 562
  Serotype 19A | 0.67 [0.61 to 0.74] | 1.13 [1.01 to 1.26]
  Serotype 19F: number analyzed (Participants) | 566 | 562
  Serotype 19F | 2.21 [2.04 to 2.40] | 3.06 [2.80 to 3.34]
  Serotype 23F: number analyzed (Participants) | 566 | 562
  Serotype 23F | 0.13 [0.12 to 0.15] | 0.25 [0.22 to 0.28]
  Serotype 8: number analyzed (Participants) | 567 | 561
  Serotype 8 | 1.62 [1.51 to 1.74] | 0.02 [0.02 to 0.02]
  Serotype 10A | 0.16 [0.14 to 0.18] | 0.02 [0.02 to 0.02]
  Serotype 11A | 1.62 [1.50 to 1.75] | 0.02 [0.02 to 0.02]
  Serotype 12F | 0.15 [0.13 to 0.17] | 0.01 [0.01 to 0.01]
  Serotype 15B: number analyzed (Participants) | 566 | 562
  Serotype 15B | 3.33 [3.00 to 3.70] | 0.04 [0.04 to 0.04]
  Serotype 22F | 2.25 [2.06 to 2.45] | 0.01 [0.01 to 0.01]
  Serotype 33F: number analyzed (Participants) | 566 | 562
  Serotype 33F | 0.31 [0.28 to 0.34] | 0.03 [0.02 to 0.03]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 1; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC to the corresponding serotype in 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (20vPnC/13vPnC) was greater than 0.5 (2-fold criterion); Geometric Mean Ratio = 0.61, 95% CI 2-sided [0.54 to 0.69] — 2-sided 95% CI was calculated by exponentiating the CI (based on the Student's t distribution) for the mean difference of the logarithm of the concentrations
Statistical Analysis 2: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.71, 95% CI 2-sided [0.64 to 0.79] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.60, 95% CI 2-sided [0.52 to 0.69] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 5; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.60, 95% CI 2-sided [0.52 to 0.70] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 6A; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.54, 95% CI 2-sided [0.45 to 0.65] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.51, 95% CI 2-sided [0.43 to 0.61] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 7: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.72, 95% CI 2-sided [0.64 to 0.80] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 8: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.59, 95% CI 2-sided [0.50 to 0.69] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 9: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 14; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.82, 95% CI 2-sided [0.70 to 0.96] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 10: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.79, 95% CI 2-sided [0.67 to 0.92] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 11: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.59, 95% CI 2-sided [0.51 to 0.69] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 12: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.72, 95% CI 2-sided [0.64 to 0.82] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 13: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.52, 95% CI 2-sided [0.44 to 0.62] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 14: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 8; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results are from serotype 6B (13vPnC serotype with the lowest GMC, not including serotype 3) in the 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (20vPnC/lowest 13vPnC) was greater than 0.5 (2-fold criterion); Geometric Mean Ratio = 26.55, 95% CI 2-sided [22.98 to 30.67] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 15: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 10A; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 14]; Geometric Mean Ratio = 2.67, 95% CI 2-sided [2.25 to 3.17] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 16: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 11A; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 14]; Geometric Mean Ratio = 26.60, 95% CI 2-sided [22.95 to 30.82] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 17: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 12F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 14]; Geometric Mean Ratio = 2.48, 95% CI 2-sided [2.08 to 2.97] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 18: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 15B; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 14]; Geometric Mean Ratio = 54.60, 95% CI 2-sided [46.35 to 64.30] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 19: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 22F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 14]; Geometric Mean Ratio = 36.80, 95% CI 2-sided [31.57 to 42.89] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 20: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 33F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 14]; Geometric Mean Ratio = 5.03, 95% CI 2-sided [4.27 to 5.92] — [estimate comment as in outcome 12, analysis 1]

13. Primary Outcome: GMC of Serotype-specific Pneumococcal IgG Antibody 1 Month After Dose 3: Primary Study Population
Description: Pneumococcal serotype-specific IgG concentrations were measured for serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 7 additional serotype: 8, 10A, 11A, 12F, 15B, 22F,33F. GMC and corresponding 2-sided 95% CI were calculated by exponentiating mean logarithm of concentrations and corresponding 2-sided 95% CI (based on Student's t distribution). Assay result below LLOQ were set to 0.5*LLOQ. GMRs were reported in statistical analysis section and were calculated by exponentiating mean difference of logarithm of concentration and corresponding 2-sided 95% CI (based on Student's t distribution).
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population (EIP)=eligible participants 42-112 days of age at first vaccination, received all 3 dose as randomized with 335-386 day of age at Dose 3 at least 1 valid immunogenicity results within 27-56 days after Dose 3, no major protocol deviation "Number of Participants Analyzed"=participants in Dose 3 EIP; "Number Analyzed"=participants with valid IgG results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per millilitre (mcg/mL)
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 497 | 504
Microgram per millilitre (mcg/mL)
  Serotype 1: number analyzed (Participants) | 494 | 502
  Serotype 1 | 1.71 [1.58 to 1.84] | 2.53 [2.33 to 2.75]
  Serotype 3: number analyzed (Participants) | 494 | 502
  Serotype 3 | 0.72 [0.67 to 0.78] | 1.09 [1.01 to 1.17]
  Serotype 4: number analyzed (Participants) | 494 | 502
  Serotype 4 | 4.11 [3.77 to 4.48] | 5.36 [4.91 to 5.85]
  Serotype 5: number analyzed (Participants) | 494 | 502
  Serotype 5 | 1.74 [1.60 to 1.89] | 2.41 [2.21 to 2.64]
  Serotype 6A: number analyzed (Participants) | 494 | 501
  Serotype 6A | 7.75 [7.04 to 8.53] | 11.82 [10.66 to 13.11]
  Serotype 6B: number analyzed (Participants) | 494 | 501
  Serotype 6B | 2.64 [2.36 to 2.95] | 4.63 [4.09 to 5.25]
  Serotype 7F: number analyzed (Participants) | 494 | 502
  Serotype 7F | 3.61 [3.40 to 3.84] | 4.93 [4.63 to 5.24]
  Serotype 9V: number analyzed (Participants) | 494 | 502
  Serotype 9V | 3.68 [3.42 to 3.97] | 5.04 [4.67 to 5.43]
  Serotype 14: number analyzed (Participants) | 493 | 501
  Serotype 14 | 4.52 [4.08 to 5.00] | 5.66 [5.12 to 6.26]
  Serotype 18C: number analyzed (Participants) | 494 | 502
  Serotype 18C | 2.71 [2.52 to 2.93] | 3.61 [3.33 to 3.91]
  Serotype 19A: number analyzed (Participants) | 494 | 502
  Serotype 19A | 4.51 [4.11 to 4.94] | 5.49 [5.02 to 6.01]
  Serotype 19F: number analyzed (Participants) | 494 | 502
  Serotype 19F | 6.19 [5.68 to 6.75] | 8.08 [7.40 to 8.83]
  Serotype 23F: number analyzed (Participants) | 494 | 502
  Serotype 23F | 2.64 [2.40 to 2.91] | 4.40 [3.95 to 4.90]
  Serotype 8: number analyzed (Participants) | 495 | 501
  Serotype 8 | 3.57 [3.32 to 3.83] | 0.03 [0.03 to 0.03]
  Serotype 10A: number analyzed (Participants) | 495 | 502
  Serotype 10A | 4.86 [4.41 to 5.36] | 0.01 [0.01 to 0.01]
  Serotype 11A: number analyzed (Participants) | 495 | 502
  Serotype 11A | 3.74 [3.44 to 4.07] | 0.02 [0.01 to 0.02]
  Serotype 12F: number analyzed (Participants) | 495 | 502
  Serotype 12F | 1.86 [1.71 to 2.01] | 0.01 [0.01 to 0.01]
  Serotype 15B: number analyzed (Participants) | 495 | 502
  Serotype 15B | 13.09 [12.10 to 14.15] | 0.02 [0.02 to 0.03]
  Serotype 22F: number analyzed (Participants) | 495 | 502
  Serotype 22F | 9.27 [8.52 to 10.08] | 0.00 [0.00 to 0.00]
  Serotype 33F: number analyzed (Participants) | 495 | 501
  Serotype 33F | 6.37 [5.83 to 6.95] | 0.01 [0.01 to 0.01]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 1; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.67, 95% CI 2-sided [0.60 to 0.75] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.66, 95% CI 2-sided [0.59 to 0.73] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.68 to 0.87] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 5; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.72, 95% CI 2-sided [0.64 to 0.81] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 6A; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.66, 95% CI 2-sided [0.57 to 0.75] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.57, 95% CI 2-sided [0.48 to 0.67] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 7: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.73, 95% CI 2-sided [0.67 to 0.80] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 8: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.73, 95% CI 2-sided [0.66 to 0.81] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 9: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 14; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.80, 95% CI 2-sided [0.69 to 0.92] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 10: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.75, 95% CI 2-sided [0.67 to 0.84] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 11: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.82, 95% CI 2-sided [0.72 to 0.93] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 12: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.68 to 0.87] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 13: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 12, analysis 1]; Geometric Mean Ratio = 0.60, 95% CI 2-sided [0.52 to 0.69] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 14: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 8; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results are from serotype 5 (13vPnC serotype with the lowest GMC, not including serotype 3) in the 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (20vPnC/lowest 13vPnC) was greater than 0.5 (2-fold criterion); Geometric Mean Ratio = 1.48, 95% CI 2-sided [1.32 to 1.66] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 15: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 10A; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Geometric Mean Ratio = 2.02, 95% CI 2-sided [1.77 to 2.30] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 16: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 11A; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Geometric Mean Ratio = 1.55, 95% CI 2-sided [1.37 to 1.75] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 17: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 12F; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.68 to 0.87] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 18: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 15B; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Geometric Mean Ratio = 5.42, 95% CI 2-sided [4.82 to 6.10] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 19: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 22F; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Geometric Mean Ratio = 3.84, 95% CI 2-sided [3.40 to 4.34] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 20: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 33F; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; Geometric Mean Ratio = 2.64, 95% CI 2-sided [2.33 to 2.99] — [estimate comment as in outcome 12, analysis 1]

14. Primary Outcome: Percentage of Participants With Predefined Antibody Levels for Concomitant Vaccine Antigens 1 Month After Dose 3: Primary Study Population
Description: Diphtheria and tetanus toxoids: concentration of antibody (AB) (in international units [IU]) to diphtheria & tetanus toxoid (prespecified level>=0.1 IU/mL); Pertussis antigens-pertussis toxin (PT), filamentous hemagglutinin (FHA), pertactin (PRN): prespecified level >=observed Anti pertussis Antibody concentration achieved by 95% of 13vPnC recipient; HBsAg prespecified level >=10 milli-IU per mL (mIU/mL); Poliovirus strains (types 1, 2 and 3): prespecified level: >=1:8; Hemophilus influenzae type b(Hib): prespecified level >=0.15 microgram per millilitre (mcg/mL) polyribosylribitol phosphate (anti-PRP) in mcg/mL. Concomitant vaccine response was assessed from subset of randomly selected study participants.
Time Frame: 1 month after Dose 3
Population: Dose 3 EIP = eligible participants 42-112 days of age at first vaccination, received all 3 doses as randomized with 335-386 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. "Number of Participants Analyzed"= participants in Dose 3 EIP and "Number Analyzed"= participants with valid assay results for specified concomitant vaccine antigen.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 497 | 504
Percentage of participants
  Diphtheria toxoid: number analyzed (Participants) | 494 | 498
  Diphtheria toxoid | 99.6 [98.5 to 100.0] | 99.8 [98.9 to 100.0]
  Tetanus toxoid: number analyzed (Participants) | 494 | 498
  Tetanus toxoid | 99.4 [98.2 to 99.9] | 100.0 [99.3 to 100.0]
  Pertussis: PT: number analyzed (Participants) | 494 | 498
  Pertussis: PT | 92.9 [90.3 to 95.0] | 95.2 [92.9 to 96.9]
  Pertussis: FHA: number analyzed (Participants) | 494 | 498
  Pertussis: FHA | 95.3 [93.1 to 97.0] | 95.2 [92.9 to 96.9]
  Pertussis: PRN: number analyzed (Participants) | 494 | 498
  Pertussis: PRN | 96.8 [94.8 to 98.1] | 95.2 [92.9 to 96.9]
  Hepatitis B: number analyzed (Participants) | 173 | 178
  Hepatitis B | 100.0 [97.9 to 100.0] | 98.9 [96.0 to 99.9]
  Poliovirus: Type 1: number analyzed (Participants) | 81 | 89
  Poliovirus: Type 1 | 100.0 [95.5 to 100.0] | 100.0 [95.9 to 100.0]
  Poliovirus: Type 2: number analyzed (Participants) | 81 | 89
  Poliovirus: Type 2 | 100.0 [95.5 to 100.0] | 100.0 [95.9 to 100.0]
  Poliovirus: Type 3: number analyzed (Participants) | 81 | 89
  Poliovirus: Type 3 | 100.0 [95.5 to 100.0] | 100.0 [95.9 to 100.0]
  Hemophilus influenzae type b: number analyzed (Participants) | 185 | 169
  Hemophilus influenzae type b | 100.0 [98.0 to 100.0] | 100.0 [97.8 to 100.0]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Diphtheria; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CIs for the percentage differences (20vPnC -13vPnC) was greater than -10%; Percent difference = -0.2, 95% CI 2-sided [-1.3 to 0.8] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions (20vPnc - 13vPnC) expressed as a percentage
Statistical Analysis 2: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Tetanus; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CIs for the percentage differences (20vPnC-13vPnC) was greater than -10%; Percent difference = -0.6, 95% CI 2-sided [-1.8 to 0.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; PT; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 2]; Percent difference = -2.3, 95% CI 2-sided [-5.3 to 0.7] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 4: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; FHA; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 2]; Percent difference = 0.2, 95% CI 2-sided [-2.6 to 2.9] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 5: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; PRN; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 2]; Percent difference = 1.6, 95% CI 2-sided [-0.9 to 4.2] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 6: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Hepatitis B; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 2]; Percent difference = 1.1, 95% CI 2-sided [-1.1 to 4.0] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Poliovirus Type 1; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Percent difference = 0.0, 95% CI 2-sided [-4.6 to 4.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Poliovirus Type 2; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 2]; Percent difference = 0.0, 95% CI 2-sided [-4.6 to 4.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Poliovirus Type 3; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 2]; Percent difference = 0.0, 95% CI 2-sided [-4.6 to 4.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Hib; Test type: Non-Inferiority — [test comment as in outcome 14, analysis 2]; Percent difference = 0.0, 95% CI 2-sided [-2.0 to 2.2] — [estimate comment as in outcome 14, analysis 1]

15. Primary Outcome: GMC of Measles Virus Antibody 1 Month After Dose 3: Primary Study Population
Description: Pre-specified vaccine antigen (measles) was administered concomitantly with 20vPnC or 13vPnC at Dose 3 and responses were measured 1 month after Dose 3. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis. GMCs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student's t distribution). The immune responses were only measured on random subset of participants.
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-112 days of age at first vaccination, received all 3 doses as randomized with 335-386 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. Here, "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population, received measles vaccine and had valid assay results for measle vaccine antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary units per millilitre
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 128 | 132
Arbitrary units per millilitre | 228.63 (186.34) [186.34 to 280.52] | 216.72 (174.92) [174.92 to 268.52]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Measles; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (20vPnC/13vPnC) was greater than 0.5 (2-fold criterion); Geometric Mean Ratio = 1.05, 95% CI 2-sided [0.79 to 1.42] — GMR and 2-sided 95% CIs were calculated by exponentiating the mean differences of the logarithms of the concentrations (20vPnC - 13vPnC) and the corresponding CIs (based on the Student's t distribution)

16. Primary Outcome: GMC of Mumps Virus Antibody 1 Month After Dose 3: Primary Study Population
Description: Pre-specified vaccine antigen (mumps) was administered concomitantly with 20vPnC or 13vPnC at Dose 3 and responses were measured 1 month after Dose 3. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis. GMCs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student's t distribution). The immune responses were only measured on random subset of participants.
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-112 days of age at first vaccination, received all 3 doses as randomized with 335-386 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. Here, "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population, received mumps vaccine and had valid assay results for mumps vaccine antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary units per millilitre
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 128 | 133
Arbitrary units per millilitre | 36.81 (29.12) [29.12 to 46.54] | 35.25 (28.14) [28.14 to 44.17]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Mumps; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Geometric Mean Ratio = 1.04, 95% CI 2-sided [0.76 to 1.44] — [estimate comment as in outcome 15, analysis 1]

17. Primary Outcome: GMC of Rubella Virus Antibody 1 Month After Dose 3: Primary Study Population
Description: Pre-specified vaccine antigen (rubella) was administered concomitantly with 20vPnC or 13vPnC at Dose 3 and responses were measured 1 month after Dose 3. Assay results below LLOQ were set to 0.5*LLOQ in the analysis. GMCs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student's t distribution). The immune responses were only measured on random subset of participants.
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-112 days of age at first vaccination, received all 3 doses as randomized with 335-386 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. Here, "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population, received rubella vaccine and had valid assay results for rubella vaccine antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: International units per millilitre
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 128 | 132
International units per millilitre | 31.81 (25.54) [25.54 to 39.62] | 38.20 (32.10) [32.10 to 45.45]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Rubella; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Geometric Mean Ratio = 0.83, 95% CI 2-sided [0.63 to 1.10] — [estimate comment as in outcome 15, analysis 1]

18. Primary Outcome: GMC of Varicella Virus Antibody 1 Month After Dose 3: Primary Study Population
Description: Pre-specified vaccine antigen (varicella) was administered concomitantly with 20vPnC or 13vPnC at Dose 3 and responses were measured 1 month after Dose 3. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis. GMCs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student's t distribution). The immune responses were only measured on random subset of participants.
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-112 days of age at first vaccination, received all 3 doses as randomized with 335-386 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. Here, "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population, received varicella vaccine and had valid assay results varicella vaccine antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Milli-international units per millilitre
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 128 | 132
Milli-international units per millilitre | 195.58 (165.14) [165.14 to 231.62] | 157.60 (133.57) [133.57 to 185.95]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Varicella; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Geometric Mean Ratio = 1.24, 95% CI 2-sided [0.98 to 1.57] — [estimate comment as in outcome 15, analysis 1]

19. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 1: Russian Cohort
Description: Local reactions included redness, swelling and, pain at the injection site, recorded by parents/legal guardians of participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm. Redness and swelling were graded as mild (>0 to 2.0 cm), moderate (> 2.0 to 7.0 cm) and severe (>7.0 cm). Pain at injection site was graded as mild (hurt if gently touched example, whimpered, winced, protested, or withdrew), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after Dose 1
Population: Safety analysis set included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies number of participants with any e-diary data after Dose 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 24 | 27
Percentage of participants
  Redness: Mild | 4.2 (0.1) [0.1 to 21.1] | 7.4 (0.9) [0.9 to 24.3]
  Redness: Moderate | 4.2 (0.1) [0.1 to 21.1] | 3.7 (0.1) [0.1 to 19.0]
  Redness: Severe | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]
  Swelling: Mild | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]
  Swelling: Moderate | 4.2 (0.1) [0.1 to 21.1] | 0 (0.0) [0.0 to 12.8]
  Swelling: Severe | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]
  Pain at Injection Site: Mild | 8.3 (1.0) [1.0 to 27.0] | 7.4 (0.9) [0.9 to 24.3]
  Pain at Injection Site: Moderate | 0 (0.0) [0.0 to 14.2] | 3.7 (0.1) [0.1 to 19.0]
  Pain at Injection Site: Severe | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]

20. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2: Russian Cohort
Description: as for outcome 19
Time Frame: Within 7 days after Dose 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 23 | 27
Percentage of participants
  Redness: Mild | 0 (0.0) [0.0 to 14.8] | 3.7 (0.1) [0.1 to 19.0]
  Redness: Moderate | 4.3 (0.1) [0.1 to 21.9] | 0 (0.0) [0.0 to 12.8]
  Redness: Severe | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 12.8]
  Swelling: Mild | 0 (0.0) [0.0 to 14.8] | 7.4 (0.9) [0.9 to 24.3]
  Swelling: Moderate | 8.7 (1.1) [1.1 to 28.0] | 0 (0.0) [0.0 to 12.8]
  Swelling: Severe | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 12.8]
  Pain at Injection Site: Mild | 8.7 (1.1) [1.1 to 28.0] | 7.4 (0.9) [0.9 to 24.3]
  Pain at Injection Site: Moderate | 4.3 (0.1) [0.1 to 21.9] | 0 (0.0) [0.0 to 12.8]
  Pain at Injection Site: Severe | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 12.8]

21. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3: Russian Cohort
Description: as for outcome 19
Time Frame: Within 7 days after Dose 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 22 | 25
Percentage of participants
  Redness: Mild | 0 [0.0 to 15.4] | 4.0 [0.1 to 20.4]
  Redness: Moderate | 4.5 [0.1 to 22.8] | 0 [0.0 to 13.7]
  Redness: Severe | 0 [0.0 to 15.4] | 4.0 [0.1 to 20.4]
  Swelling: Mild | 0 [0.0 to 15.4] | 0 [0.0 to 13.7]
  Swelling: Moderate | 9.1 [1.1 to 29.2] | 0 [0.0 to 13.7]
  Swelling: Severe | 0 [0.0 to 15.4] | 4.0 [0.1 to 20.4]
  Pain at Injection Site: Mild | 13.6 [2.9 to 34.9] | 8.0 [1.0 to 26.0]
  Pain at Injection Site: Moderate | 0 [0.0 to 15.4] | 0 [0.0 to 13.7]
  Pain at Injection Site: Severe | 0 [0.0 to 15.4] | 0 [0.0 to 13.7]

22. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1: Russian Cohort
Description: Systemic events: fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participant's using e-diary. Fever: temperature >=38.0 degree C & categorized as >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0-degree C. Decreased appetite: was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased/prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability: mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper & Pearson method.
Time Frame: Within 7 Days after Dose 1
Population: Safety analysis set: all participants who received at least 1 dose of 20vPnC or 13vPnC & had safety data assessed after any dose. Here, "Number of Participants Analyzed" signifies number of participants with any e-diary data after Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 24 | 27
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 4.2 (0.1) [0.1 to 21.1] | 0 (0.0) [0.0 to 12.8]
  Fever: >38.4 degrees C to 38.9 degrees C | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]
  Fever: >38.9 degrees C to 40.0 degrees C | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]
  Fever: >40.0 degrees C | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]
  Decreased appetite: Mild | 16.7 (4.7) [4.7 to 37.4] | 14.8 (4.2) [4.2 to 33.7]
  Decreased appetite: Moderate | 0 (0.0) [0.0 to 14.2] | 3.7 (0.1) [0.1 to 19.0]
  Decreased appetite: Severe | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]
  Drowsiness: Mild | 20.8 (7.1) [7.1 to 42.2] | 18.5 (6.3) [6.3 to 38.1]
  Drowsiness: Moderate | 8.3 (1.0) [1.0 to 27.0] | 11.1 (2.4) [2.4 to 29.2]
  Drowsiness: Severe | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 12.8]
  Irritability: Mild | 12.5 (2.7) [2.7 to 32.4] | 7.4 (0.9) [0.9 to 24.3]
  Irritability: Moderate | 8.3 (1.0) [1.0 to 27.0] | 14.8 (4.2) [4.2 to 33.7]
  Irritability: Severe | 4.2 (0.1) [0.1 to 21.1] | 0 (0.0) [0.0 to 12.8]

23. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2: Russian Cohort
Description: Systemic events: fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participants using an e-diary. Fever: temperature >=38.0 degree C and categorized as >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0-degree C. Decreased appetite: mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased/prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability: mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper & Pearson method.
Time Frame: Within 7 Days after Dose 2
Population: Safety analysis set: all participants who received at least 1 dose of 20vPnC or 13vPnC & had safety data assessed after any dose. Here," Number of Participants Analyzed": number of participants with any e-diary data after Dose 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 23 | 27
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 0 (0.0) [0.0 to 14.8] | 11.1 (2.4) [2.4 to 29.2]
  Fever: >38.4 degrees C to 38.9 degrees C | 4.3 (0.1) [0.1 to 21.9] | 0 (0.0) [0.0 to 12.8]
  Fever: >38.9 degrees C to 40.0 degrees C | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 12.8]
  Fever: >40.0 degrees C | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 12.8]
  Decreased appetite: Mild | 4.3 (0.1) [0.1 to 21.9] | 7.4 (0.9) [0.9 to 24.3]
  Decreased appetite: Moderate | 4.3 (0.1) [0.1 to 21.9] | 3.7 (0.1) [0.1 to 19.0]
  Decreased appetite: Severe | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 12.8]
  Drowsiness: Mild | 4.3 (0.1) [0.1 to 21.9] | 3.7 (0.1) [0.1 to 19.0]
  Drowsiness: Moderate | 0 (0.0) [0.0 to 14.8] | 3.7 (0.1) [0.1 to 19.0]
  Drowsiness: Severe | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 12.8]
  Irritability: Mild | 13.0 (2.8) [2.8 to 33.6] | 22.2 (8.6) [8.6 to 42.3]
  Irritability: Moderate | 4.3 (0.1) [0.1 to 21.9] | 18.5 (6.3) [6.3 to 38.1]
  Irritability: Severe | 0 (0.0) [0.0 to 14.8] | 3.7 (0.1) [0.1 to 19.0]

24. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3: Russian Cohort
Description: as for outcome 23
Time Frame: Within 7 Days after Dose 3
Population: Safety analysis set: all participants who received at least 1 dose of 20vPnC or 13vPnC & had safety data assessed after any dose. Here," Number of Participants Analyzed": number of participants with any e-diary data after Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 22 | 25
Percentage of participants
  Fever: >=38.0 degrees C to 38.4 degrees C | 0 (0.0) [0.0 to 15.4] | 0 (0.0) [0.0 to 13.7]
  Fever: >38.4 degrees C to 38.9 degrees C | 0 (0.0) [0.0 to 15.4] | 4.0 (0.1) [0.1 to 20.4]
  Fever: >38.9 degrees C to 40.0 degrees C | 4.5 (0.1) [0.1 to 22.8] | 0 (0.0) [0.0 to 13.7]
  Fever: >40.0 degrees C | 0 (0.0) [0.0 to 15.4] | 0 (0.0) [0.0 to 13.7]
  Decreased appetite: Mild | 9.1 (1.1) [1.1 to 29.2] | 8.0 (1.0) [1.0 to 26.0]
  Decreased appetite: Moderate | 9.1 (1.1) [1.1 to 29.2] | 0 (0.0) [0.0 to 13.7]
  Decreased appetite: Severe | 0 (0.0) [0.0 to 15.4] | 0 (0.0) [0.0 to 13.7]
  Drowsiness: Mild | 13.6 (2.9) [2.9 to 34.9] | 20.0 (6.8) [6.8 to 40.7]
  Drowsiness: Moderate | 0 (0.0) [0.0 to 15.4] | 4.0 (0.1) [0.1 to 20.4]
  Drowsiness: Severe | 0 (0.0) [0.0 to 15.4] | 0 (0.0) [0.0 to 13.7]
  Irritability: Mild | 27.3 (10.7) [10.7 to 50.2] | 16.0 (4.5) [4.5 to 36.1]
  Irritability: Moderate | 9.1 (1.1) [1.1 to 29.2] | 8.0 (1.0) [1.0 to 26.0]
  Irritability: Severe | 0 (0.0) [0.0 to 15.4] | 0 (0.0) [0.0 to 13.7]

25. Primary Outcome: Percentage of Participants With AEs From Dose 1 to 1 Month After Dose 2: Russian Cohort
Description: as for outcome 7
Time Frame: From Dose 1 to 1 month after Dose 2
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 24 | 27
Percentage of participants | 8.3 (1.0) [1.0 to 27.0] | 3.7 (0.1) [0.1 to 19.0]

26. Primary Outcome: Percentage of Participants With AEs From Dose 3 to 1 Month After Dose 3: Russian Cohort
Description: An AE was any untoward medical occurrence in a participants, temporally associated with the use of study treatment, whether or not considered related to the study treatment. 95% CI was based on the Clopper and Pearson method. AEs reported in this outcome measure excluded local reactions and systemic events collected from an e-diary.
Time Frame: From Dose 3 to 1 month after Dose 3
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 22 | 25
Percentage of participants | 4.5 (0.1) [0.1 to 22.8] | 0 (0.0) [0.0 to 13.7]

27. Primary Outcome: Percentage of Participants With SAEs From Dose 1 to 1 Month After Dose 3: Russian Cohort
Description: as for outcome 9
Time Frame: From Dose 1 to 1 month after Dose 3
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 24 | 27
Percentage of participants | 0 [0 to 14.2] | 0 [0 to 12.8]

28. Primary Outcome: Percentage of Participants With NDCMC From Dose 1 to 1 Month After Dose 3: Russian Cohort
Description: as for outcome 10
Time Frame: From Dose 1 to 1 month after Dose 3
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 24 | 27
Percentage of participants | 0 [0 to 14.2] | 0 [0 to 12.8]

29. Primary Outcome: Percentage of Participants With Predefined Pneumococcal IgG Antibody 1 Month After Dose 2: Russian Cohort
Description: Predefined IgG concentrations were as follows: for serotype 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, 33F: >=0.35 mcg/mL, for serotype 5: >=0.23 mcg/mL, for serotype 6B. >=0.10 mcg/mL and for serotype 19A: >=0.12 mcg/mL. 95% CI was based on the Clopper and Pearson method.
Time Frame: 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population: eligible participants 42-70 days of age at first vaccination, received first 2 doses as randomized, at least 1 valid immunogenicity results within 27 to 56 days after Dose 2, no other major protocol deviations. "Number of Participants Analyzed"= participants in Dose 2 evaluable immunogenicity population; "Number Analyzed"= participants with valid IgG results for specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 24 | 27
Percentage of participants
  Serotype 1 | 70.8 (48.9) [48.9 to 87.4] | 77.8 (57.7) [57.7 to 91.4]
  Serotype 3 | 37.5 (18.8) [18.8 to 59.4] | 59.3 (38.8) [38.8 to 77.6]
  Serotype 4 | 75.0 (53.3) [53.3 to 90.2] | 74.1 (53.7) [53.7 to 88.9]
  Serotype 5 | 66.7 (44.7) [44.7 to 84.4] | 81.5 (61.9) [61.9 to 93.7]
  Serotype 6A | 54.2 (32.8) [32.8 to 74.4] | 81.5 (61.9) [61.9 to 93.7]
  Serotype 6B | 20.8 (7.1) [7.1 to 42.2] | 59.3 (38.8) [38.8 to 77.6]
  Serotype 7F | 95.8 (78.9) [78.9 to 99.9] | 92.6 (75.7) [75.7 to 99.1]
  Serotype 9V | 41.7 (22.1) [22.1 to 63.4] | 81.5 (61.9) [61.9 to 93.7]
  Serotype 14 | 83.3 (62.6) [62.6 to 95.3] | 85.2 (66.3) [66.3 to 95.8]
  Serotype 18C | 66.7 (44.7) [44.7 to 84.4] | 81.5 (61.9) [61.9 to 93.7]
  Serotype 19A | 87.5 (67.6) [67.6 to 97.3] | 92.6 (75.7) [75.7 to 99.1]
  Serotype 19F | 79.2 (57.8) [57.8 to 92.9] | 96.3 (81.0) [81.0 to 99.9]
  Serotype 23F | 37.5 (18.8) [18.8 to 59.4] | 70.4 (49.8) [49.8 to 86.2]
  Serotype 8 | 75.0 (53.3) [53.3 to 90.2] | 33.3 (16.5) [16.5 to 54.0]
  Serotype 10A | 41.7 (22.1) [22.1 to 63.4] | 18.5 (6.3) [6.3 to 38.1]
  Serotype 11A | 83.3 (62.6) [62.6 to 95.3] | 18.5 (6.3) [6.3 to 38.1]
  Serotype 12F | 12.5 (2.7) [2.7 to 32.4] | 14.8 (4.2) [4.2 to 33.7]
  Serotype 15B | 66.7 (44.7) [44.7 to 84.4] | 33.3 (16.5) [16.5 to 54.0]
  Serotype 22F | 66.7 (44.7) [44.7 to 84.4] | 14.8 (4.2) [4.2 to 33.7]
  Serotype 33F | 45.8 (25.6) [25.6 to 67.2] | 25.9 (11.1) [11.1 to 46.3]

30. Primary Outcome: GMC of Serotype-specific Pneumococcal IgG Antibody 1 Month After Dose 2: Russian Cohort
Description: Pneumococcal serotype-specific IgG concentrations were measured for serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F and 7 additional serotypes: 8, 10A, 11A, 12F, 15B, 22F, 33F. Assay results below the LLOQ were set to 0.5 * LLOQ. GMC and corresponding 2-sided 95% CIs were calculated by exponentiating mean logarithm of concentration, and the corresponding 2-sided 95% CIs (based on Student's t distribution).
Time Frame: 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population: eligible participants 42-70days of age at first vaccination, received first 2 doses as randomized, at least 1 valid immunogenicity results within 27 to 56 days after Dose 2, no other major protocol deviations. "Number of Participants Analyzed"= Participants in Dose 2 evaluable immunogenicity population; "Number Analyzed"= participants with valid IgG results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per millilitre (mcg/mL)
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 24 | 27
Microgram per millilitre (mcg/mL)
  Serotype 1 | 0.76 (0.49) [0.49 to 1.19] | 1.04 (0.64) [0.64 to 1.69]
  Serotype 3 | 0.28 (0.19) [0.19 to 0.42] | 0.47 (0.31) [0.31 to 0.72]
  Serotype 4 | 0.67 (0.45) [0.45 to 1.00] | 1.00 (0.58) [0.58 to 1.71]
  Serotype 5 | 0.53 (0.31) [0.31 to 0.92] | 0.75 (0.40) [0.40 to 1.40]
  Serotype 6A | 0.45 (0.20) [0.20 to 1.03] | 1.57 (0.80) [0.80 to 3.10]
  Serotype 6B | 0.07 (0.03) [0.03 to 0.16] | 0.27 (0.12) [0.12 to 0.63]
  Serotype 7F | 1.06 (0.68) [0.68 to 1.65] | 1.89 (1.32) [1.32 to 2.71]
  Serotype 9V | 0.44 (0.23) [0.23 to 0.84] | 1.22 (0.73) [0.73 to 2.06]
  Serotype 14 | 1.56 (0.88) [0.88 to 2.75] | 2.66 (1.46) [1.46 to 4.86]
  Serotype 18C | 0.94 (0.46) [0.46 to 1.91] | 0.94 (0.50) [0.50 to 1.78]
  Serotype 19A | 1.15 (0.47) [0.47 to 2.82] | 1.21 (0.59) [0.59 to 2.49]
  Serotype 19F | 1.51 (0.84) [0.84 to 2.72] | 3.32 (2.03) [2.03 to 5.44]
  Serotype 23F | 0.25 (0.11) [0.11 to 0.55] | 0.73 (0.37) [0.37 to 1.42]
  Serotype 8 | 0.79 (0.37) [0.37 to 1.69] | 0.07 (0.03) [0.03 to 0.18]
  Serotype 10A | 0.31 (0.10) [0.10 to 0.94] | 0.04 (0.01) [0.01 to 0.10]
  Serotype 11A | 0.83 (0.43) [0.43 to 1.60] | 0.04 (0.02) [0.02 to 0.09]
  Serotype 12F | 0.06 (0.03) [0.03 to 0.11] | 0.02 (0.01) [0.01 to 0.04]
  Serotype 15B | 1.19 (0.46) [0.46 to 3.05] | 0.16 (0.05) [0.05 to 0.50]
  Serotype 22F | 0.48 (0.16) [0.16 to 1.47] | 0.02 (0.01) [0.01 to 0.06]
  Serotype 33F | 0.40 (0.18) [0.18 to 0.88] | 0.07 (0.03) [0.03 to 0.16]

31. Primary Outcome: GMC of Serotype-specific Pneumococcal IgG Antibody 1 Month After Dose 3: Russian Cohort
Description: Pneumococcal serotype-specific IgG concentrations were measured for serum samples for 13vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F and additional serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. Assay results below the LLOQ were set to 0.5 * LLOQ. GMC and corresponding 2-sided 95% CIs were calculated by exponentiating mean logarithm of concentration, and the corresponding 2-sided 95% CIs (based on Student's t distribution).
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-70 days of age at first vaccination, received all 3 doses as randomized with 335-455 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. Here, "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population; "Number Analyzed"= participants with valid IgG results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per millilitre (mcg/mL)
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 22 | 24
Microgram per millilitre (mcg/mL)
  Serotype 1 | 1.61 (0.93) [0.93 to 2.78] | 1.65 (0.94) [0.94 to 2.90]
  Serotype 3 | 0.84 (0.44) [0.44 to 1.60] | 0.57 (0.32) [0.32 to 1.01]
  Serotype 4 | 3.05 (1.50) [1.50 to 6.20] | 3.04 (1.72) [1.72 to 5.36]
  Serotype 5 | 1.50 (0.80) [0.80 to 2.82] | 1.72 (0.90) [0.90 to 3.29]
  Serotype 6A | 6.63 (2.96) [2.96 to 14.86] | 5.63 (2.96) [2.96 to 10.72]
  Serotype 6B | 1.94 (0.82) [0.82 to 4.56] | 1.49 (0.67) [0.67 to 3.32]
  Serotype 7F | 3.53 (1.97) [1.97 to 6.33] | 4.14 (2.73) [2.73 to 6.26]
  Serotype 9V | 2.32 (1.28) [1.28 to 4.19] | 2.27 (1.19) [1.19 to 4.35]
  Serotype 14 | 4.01 (1.64) [1.64 to 9.77] | 5.06 (3.04) [3.04 to 8.40]
  Serotype 18C | 2.60 (1.24) [1.24 to 5.44] | 2.64 (1.49) [1.49 to 4.69]
  Serotype 19A | 4.81 (2.07) [2.07 to 11.16] | 2.69 (1.12) [1.12 to 6.45]
  Serotype 19F | 4.97 (2.30) [2.30 to 10.76] | 4.58 (2.36) [2.36 to 8.90]
  Serotype 23F | 3.52 (1.68) [1.68 to 7.38] | 2.96 (1.33) [1.33 to 6.56]
  Serotype 8 | 1.33 (0.50) [0.50 to 3.56] | 0.09 (0.04) [0.04 to 0.24]
  Serotype 10A | 1.99 (0.63) [0.63 to 6.29] | 0.03 (0.01) [0.01 to 0.09]
  Serotype 11A | 1.50 (0.58) [0.58 to 3.87] | 0.06 (0.02) [0.02 to 0.16]
  Serotype 12F | 0.17 (0.05) [0.05 to 0.56] | 0.02 (0.01) [0.01 to 0.03]
  Serotype 15B | 4.90 (1.67) [1.67 to 14.37] | 0.07 (0.03) [0.03 to 0.20]
  Serotype 22F | 1.52 (0.38) [0.38 to 6.03] | 0.02 (0.01) [0.01 to 0.08]
  Serotype 33F | 1.38 (0.53) [0.53 to 3.59] | 0.04 (0.02) [0.02 to 0.10]

32. Secondary Outcome: Percentage of Participants With Predefined Pneumococcal IgG Antibody 1 Month After Dose 3: Primary Study Population
Description: Predefined IgG concentrations were as follows: for serotype 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, 33F: >=0.35 mcg/mL, for serotype 5: >=0.23 mcg/mL, for serotype 6B: >=0.10 mcg/mL and for serotype 19A: >=0.12 mcg/mL. 95% CI was based on the Clopper and Pearson method.
Time Frame: 1 Month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-112 days of age at first vaccination, received all 3 doses as randomized with 335-386 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population; "Number Analyzed"= participants with valid IgG results for specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 497 | 504
Percentage of participants
  Serotype 1: number analyzed (Participants) | 494 | 502
  Serotype 1 | 97.2 [95.3 to 98.4] | 98.2 [96.6 to 99.2]
  Serotype 3: number analyzed (Participants) | 494 | 502
  Serotype 3 | 82.6 [79.0 to 85.8] | 93.2 [90.7 to 95.3]
  Serotype 4: number analyzed (Participants) | 494 | 502
  Serotype 4 | 99.2 [97.9 to 99.8] | 99.2 [98.0 to 99.8]
  Serotype 5: number analyzed (Participants) | 494 | 502
  Serotype 5 | 98.4 [96.8 to 99.3] | 98.0 [96.4 to 99.0]
  Serotype 6A: number analyzed (Participants) | 494 | 501
  Serotype 6A | 98.8 [97.4 to 99.6] | 98.8 [97.4 to 99.6]
  Serotype 6B: number analyzed (Participants) | 494 | 501
  Serotype 6B | 98.4 [96.8 to 99.3] | 97.6 [95.9 to 98.8]
  Serotype 7F: number analyzed (Participants) | 494 | 502
  Serotype 7F | 99.6 [98.5 to 100.0] | 100.0 [99.3 to 100.0]
  Serotype 9V: number analyzed (Participants) | 494 | 502
  Serotype 9V | 99.2 [97.9 to 99.8] | 98.8 [97.4 to 99.6]
  Serotype 14: number analyzed (Participants) | 493 | 501
  Serotype 14 | 96.6 [94.5 to 98.0] | 98.0 [96.4 to 99.0]
  Serotype 18C: number analyzed (Participants) | 494 | 502
  Serotype 18C | 99.2 [97.9 to 99.8] | 98.2 [96.6 to 99.2]
  Serotype 19A: number analyzed (Participants) | 494 | 502
  Serotype 19A | 99.6 [98.5 to 100.0] | 99.6 [98.6 to 100.0]
  Serotype 19F: number analyzed (Participants) | 494 | 502
  Serotype 19F | 99.6 [98.5 to 100.0] | 99.4 [98.3 to 99.9]
  Serotype 23F: number analyzed (Participants) | 494 | 502
  Serotype 23F | 96.4 [94.3 to 97.8] | 97.2 [95.4 to 98.5]
  Serotype 8: number analyzed (Participants) | 495 | 501
  Serotype 8 | 99.2 [97.9 to 99.8] | 3.6 [2.1 to 5.6]
  Serotype 10A: number analyzed (Participants) | 495 | 502
  Serotype 10A | 97.8 [96.1 to 98.9] | 1.6 [0.7 to 3.1]
  Serotype 11A: number analyzed (Participants) | 495 | 502
  Serotype 11A | 98.4 [96.8 to 99.3] | 4.6 [2.9 to 6.8]
  Serotype 12F: number analyzed (Participants) | 495 | 502
  Serotype 12F | 96.6 [94.6 to 98.0] | 0.2 [0.0 to 1.1]
  Serotype 15B: number analyzed (Participants) | 495 | 502
  Serotype 15B | 99.4 [98.2 to 99.9] | 4.8 [3.1 to 7.0]
  Serotype 22F: number analyzed (Participants) | 495 | 502
  Serotype 22F | 99.2 [97.9 to 99.8] | 1.4 [0.6 to 2.9]
  Serotype 33F: number analyzed (Participants) | 495 | 501
  Serotype 33F | 98.6 [97.1 to 99.4] | 1.8 [0.8 to 3.4]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 1 \; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = -1.0, 95% CI 2-sided [-3.1 to 0.9] — 2-Sided 95% CIs are calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage
Statistical Analysis 2: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 3; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = -10.6, 95% CI 2-sided [-14.7 to -6.7] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 3: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 4; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = 0.0, 95% CI 2-sided [-1.4 to 1.3] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 4: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 5; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = 0.4, 95% CI 2-sided [-1.4 to 2.2] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 5: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 6A; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = 0.0, 95% CI 2-sided [-1.6 to 1.5] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 6: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 6B; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = 0.8, 95% CI 2-sided [-1.1 to 2.7] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 7: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 7F; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = -0.4, 95% CI 2-sided [-1.5 to 0.4] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 8: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 9V; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = 0.4, 95% CI 2-sided [-1.0 to 1.9] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 9: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 14; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = -1.5, 95% CI 2-sided [-3.7 to 0.6] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 10: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 18C; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = 1.0, 95% CI 2-sided [-0.5 to 2.7] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 11: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 19A; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = 0.0, 95% CI 2-sided [-1.1 to 1.1] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 12: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 19F; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = 0.2, 95% CI 2-sided [-0.9 to 1.4] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 13: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 23F; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group; Percent difference = -0.9, 95% CI 2-sided [-3.2 to 1.4] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 14: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 8; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results are from serotype 23F(13vPnC serotype with the lowest percentage, not including serotype 3) in the 13vPnC group; Percent difference = 2.0, 95% CI 2-sided [0.4 to 3.9] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 15: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 10A; Test type: Non-Inferiority — [test comment as in outcome 32, analysis 14]; Percent difference = 0.6, 95% CI 2-sided [-1.5 to 2.7] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 16: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 11A; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results are from serotype 23F (13vPnC serotype with the lowest percentage, not including serotype 3) in the 13vPnC group; Percent difference = 1.2, 95% CI 2-sided [-0.7 to 3.2] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 17: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 12F; Test type: Non-Inferiority — [test comment as in outcome 32, analysis 16]; Percent difference = -0.6, 95% CI 2-sided [-2.9 to 1.6] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 18: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 15B; Test type: Non-Inferiority — [test comment as in outcome 32, analysis 16]; Percent difference = 2.2, 95% CI 2-sided [0.7 to 4.1] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 19: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 22F; Test type: Non-Inferiority — [test comment as in outcome 32, analysis 14]; Percent difference = 2.0, 95% CI 2-sided [0.4 to 3.9] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage
Statistical Analysis 20: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Serotype 33F; Test type: Non-Inferiority — [test comment as in outcome 32, analysis 16]; Percent difference = 1.4, 95% CI 2-sided [-0.4 to 3.4] — 2-Sided 95% CI based on the Miettinen and Nurminen method for the difference in proportions expressed as a percentage

33. Secondary Outcome: Geometric Mean Titers (GMTs) of Serotype-specific Opsonophagocytic Activity (OPA) 1 Month After Dose 2: Primary Study Population
Description: OPA titers for the 20 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, and 33F) were determined in randomly selected subsets of participants at 1 month after Dose 2. Results were expressed as OPA titers. GMTs and 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs based on the Student's t distribution.
Time Frame: 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population: eligible participants 42-112 days of age at first vaccination, received first 2 doses as randomized, at least 1 valid immunogenicity results within 27 to 56 days after Dose 2, no other major protocol deviations. "Number of Participants Analyzed"= participants in Dose 2 evaluable immunogenicity population, "Number Analyzed"= participants with valid OPA assay results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 567 | 562
Titers
  Serotype 1: number analyzed (Participants) | 113 | 107
  Serotype 1 | 14 [12 to 16] | 23 [19 to 28]
  Serotype 3: number analyzed (Participants) | 114 | 102
  Serotype 3 | 31 [26 to 36] | 40 [34 to 47]
  Serotype 4: number analyzed (Participants) | 113 | 112
  Serotype 4 | 333 [270 to 413] | 391 [314 to 486]
  Serotype 5: number analyzed (Participants) | 112 | 102
  Serotype 5 | 21 [18 to 23] | 27 [23 to 31]
  Serotype 6A: number analyzed (Participants) | 112 | 100
  Serotype 6A | 347 [273 to 441] | 409 [318 to 527]
  Serotype 6B: number analyzed (Participants) | 106 | 97
  Serotype 6B | 54 [42 to 71] | 105 [76 to 144]
  Serotype 7F: number analyzed (Participants) | 114 | 111
  Serotype 7F | 858 [736 to 1000] | 895 [781 to 1027]
  Serotype 9V: number analyzed (Participants) | 567 | 112
  Serotype 9V | 233 [182 to 298] | 285 [228 to 358]
  Serotype 14: number analyzed (Participants) | 111 | 101
  Serotype 14 | 287 [215 to 383] | 360 [264 to 489]
  Serotype 18C: number analyzed (Participants) | 114 | 112
  Serotype 18C | 588 [467 to 741] | 719 [590 to 876]
  Serotype 19A: number analyzed (Participants) | 115 | 111
  Serotype 19A | 57 [43 to 75] | 91 [69 to 121]
  Serotype 19F: number analyzed (Participants) | 114 | 103
  Serotype 19F | 97 [81 to 116] | 117 [94 to 146]
  Serotype 23F: number analyzed (Participants) | 105 | 108
  Serotype 23F | 59 [42 to 84] | 68 [48 to 96]
  Serotype 8: number analyzed (Participants) | 103 | 115
  Serotype 8 | 164 [133 to 203] | 17 [15 to 18]
  Serotype 10A: number analyzed (Participants) | 109 | 115
  Serotype 10A | 855 [610 to 1199] | 39 [34 to 44]
  Serotype 11A: number analyzed (Participants) | 105 | 116
  Serotype 11A | 327 [253 to 423] | 49 [47 to 51]
  Serotype 12F: number analyzed (Participants) | 96 | 116
  Serotype 12F | 4788 [3779 to 6067] | 26 [23 to 28]
  Serotype 15B: number analyzed (Participants) | 104 | 117
  Serotype 15B | 846 [605 to 1183] | 17 [15 to 19]
  Serotype 22F: number analyzed (Participants) | 104 | 117
  Serotype 22F | 4444 [3666 to 5386] | 10 [9 to 11]
  Serotype 33F: number analyzed (Participants) | 102 | 115
  Serotype 33F | 2373 [1759 to 3202] | 178 [163 to 195]

34. Secondary Outcome: Geometric Mean Titers (GMTs) of Serotype-specific Opsonophagocytic Activity (OPA) 1 Month After Dose 3: Primary Study Population
Description: OPA titers for the 20 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, and 33F) were determined in randomly selected subsets of participants at 1 month after Dose 3. Results were expressed as OPA titers. GMTs and 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs based on the Student's t distribution.
Time Frame: 1 Month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-112 days of age at first vaccination, received all 3 doses as randomized with 335-386 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population; "Number Analyzed"= participants with valid assay results for specified OPA serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 497 | 504
Titers
  Serotype 1: number analyzed (Participants) | 104 | 97
  Serotype 1 | 54 [43 to 69] | 101 [79 to 129]
  Serotype 3: number analyzed (Participants) | 105 | 98
  Serotype 3 | 99 [84 to 117] | 129 [111 to 150]
  Serotype 4: number analyzed (Participants) | 99 | 100
  Serotype 4 | 904 [752 to 1086] | 992 [777 to 1266]
  Serotype 5: number analyzed (Participants) | 106 | 98
  Serotype 5 | 60 [50 to 72] | 82 [66 to 101]
  Serotype 6A: number analyzed (Participants) | 105 | 96
  Serotype 6A | 1101 [897 to 1350] | 1304 [1018 to 1671]
  Serotype 6B: number analyzed (Participants) | 102 | 96
  Serotype 6B | 537 [408 to 706] | 864 [664 to 1125]
  Serotype 7F: number analyzed (Participants) | 100 | 103
  Serotype 7F | 1811 [1553 to 2112] | 2197 [1905 to 2533]
  Serotype 9V: number analyzed (Participants) | 97 | 99
  Serotype 9V | 3254 [2596 to 4079] | 4544 [3681 to 5610]
  Serotype 14: number analyzed (Participants) | 105 | 95
  Serotype 14 | 738 [606 to 899] | 926 [751 to 1142]
  Serotype 18C: number analyzed (Participants) | 98 | 102
  Serotype 18C | 1296 [1048 to 1602] | 1870 [1489 to 2348]
  Serotype 19A: number analyzed (Participants) | 99 | 100
  Serotype 19A | 754 [627 to 907] | 707 [558 to 896]
  Serotype 19F: number analyzed (Participants) | 105 | 97
  Serotype 19F | 183 [140 to 237] | 258 [192 to 347]
  Serotype 23F: number analyzed (Participants) | 100 | 101
  Serotype 23F | 697 [530 to 917] | 975 [734 to 1296]
  Serotype 8: number analyzed (Participants) | 92 | 105
  Serotype 8 | 1398 [1088 to 1796] | 31 [25 to 39]
  Serotype 10A: number analyzed (Participants) | 91 | 107
  Serotype 10A | 3403 [2600 to 4455] | 69 [52 to 91]
  Serotype 11A: number analyzed (Participants) | 87 | 92
  Serotype 11A | 2966 [2212 to 3978] | 66 [51 to 85]
  Serotype 12F: number analyzed (Participants) | 88 | 108
  Serotype 12F | 5501 [4499 to 6725] | 29 [25 to 35]
  Serotype 15B: number analyzed (Participants) | 91 | 504
  Serotype 15B | 2676 [1948 to 3677] | 23 [18 to 30]
  Serotype 22F: number analyzed (Participants) | 83 | 103
  Serotype 22F | 6523 [4848 to 8777] | 17 [13 to 24]
  Serotype 33F: number analyzed (Participants) | 72 | 99
  Serotype 33F | 11315 [8107 to 15794] | 708 [545 to 920]

35. Secondary Outcome: Geometric Mean Fold Rise (GMFRs) of IgG Concentrations From Before Dose 3 to 1 Month After Dose 3: Primary Study Population
Description: 20vPnC serotypes included: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, and 33F. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis. GMFRs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student's t distribution).
Time Frame: Before Dose 3 to 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-112 days of age at first vaccination, received all 3 doses as randomized with 335-386 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population; "Number Analysed"= participants in Dose 3 EIP at both timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 497 | 504
Fold rise
  Serotype 1: number analyzed (Participants) | 482 | 495
  Serotype 1 | 13.9 [12.7 to 15.3] | 13.9 [12.8 to 15.1]
  Serotype 3: number analyzed (Participants) | 482 | 495
  Serotype 3 | 13.7 [12.4 to 15.1] | 15.2 [13.9 to 16.7]
  Serotype 4: number analyzed (Participants) | 482 | 495
  Serotype 4 | 29.8 [27.0 to 32.9] | 27.7 [25.0 to 30.6]
  Serotype 5: number analyzed (Participants) | 482 | 495
  Serotype 5 | 14.0 [12.9 to 15.2] | 13.6 [12.6 to 14.7]
  Serotype 6A: number analyzed (Participants) | 482 | 493
  Serotype 6A | 26.9 [24.2 to 30.0] | 28.7 [25.9 to 31.7]
  Serotype 6B: number analyzed (Participants) | 481 | 493
  Serotype 6B | 36.8 [33.3 to 40.6] | 40.2 [36.8 to 44.0]
  Serotype 7F: number analyzed (Participants) | 482 | 495
  Serotype 7F | 8.5 [7.9 to 9.2] | 9.3 [8.6 to 10.0]
  Serotype 9V: number analyzed (Participants) | 482 | 495
  Serotype 9V | 22.5 [20.4 to 24.7] | 19.9 [18.3 to 21.6]
  Serotype 14: number analyzed (Participants) | 480 | 494
  Serotype 14 | 9.7 [8.7 to 10.8] | 8.4 [7.6 to 9.4]
  Serotype 18C: number analyzed (Participants) | 482 | 495
  Serotype 18C | 15.8 [14.5 to 17.1] | 17.0 [15.7 to 18.4]
  Serotype 19A: number analyzed (Participants) | 481 | 495
  Serotype 19A | 39.3 [34.6 to 44.7] | 40.7 [36.4 to 45.5]
  Serotype 19F: number analyzed (Participants) | 482 | 495
  Serotype 19F | 20.5 [18.4 to 22.9] | 21.4 [19.4 to 23.7]
  Serotype 23F: number analyzed (Participants) | 482 | 495
  Serotype 23F | 32.3 [29.2 to 35.7] | 38.3 [34.7 to 42.4]
  Serotype 8: number analyzed (Participants) | 483 | 493
  Serotype 8 | 12.7 [11.6 to 13.9] | 1.4 [1.3 to 1.5]
  Serotype 10A: number analyzed (Participants) | 484 | 495
  Serotype 10A | 14.8 [13.3 to 16.4] | 1.1 [1.0 to 1.2]
  Serotype 11A: number analyzed (Participants) | 484 | 495
  Serotype 11A | 13.8 [12.4 to 15.3] | 1.1 [1.0 to 1.2]
  Serotype 12F: number analyzed (Participants) | 484 | 495
  Serotype 12F | 16.5 [15.0 to 18.0] | 1.0 [1.0 to 1.1]
  Serotype 15B: number analyzed (Participants) | 484 | 495
  Serotype 15B | 13.4 [11.9 to 15.1] | 1.3 [1.2 to 1.4]
  Serotype 22F: number analyzed (Participants) | 484 | 495
  Serotype 22F | 12.8 [11.5 to 14.3] | 1.3 [1.1 to 1.4]
  Serotype 33F: number analyzed (Participants) | 484 | 494
  Serotype 33F | 12.9 [11.6 to 14.3] | 1.1 [1.0 to 1.2]

36. Secondary Outcome: Percentage of Participants With Predefined Antibody Levels for Concomitant Vaccine Antigens 1 Month After Dose 2: Primary Study Population
Description: Pre-specified vaccines were administered concomitantly with 20vPnC or 13vPnC and responses assessed using pre-defined levels as follows: Diphtheria and tetanus toxoids: concentration of antibody (in international units [IU]) to diphtheria and tetanus toxoid (prespecified level >= observed anti-pertussis antibody concentration achieved by 95% of 13vPnC recipients); Poliomyelitis: NA titers to poliovirus types 1, 2, and 3 (prespecified level NA titer >=1:8); and Hib: concentration of antibody to Hib (PRP) in mcg/mL (prespecified level >=0.15 mcg/mL anti-PRP). 2-sided 95% CI was based on Clopper and Pearson method. The assays were performed on randomly selected subsets.
Time Frame: 1 month after Dose 2
Population: Dose 2 EIP=eligible participants 42-112 days of age at first vaccine, received 2 dose as randomized, at least 1 valid immunogenicity result from blood collection (27 to 56 days after Dose 2), no other major protocol deviations. "Number of Participants Analyzed"= participants in Dose 2 evaluable immunogenicity population; "Number Analyzed"= participants with valid assay results for specified concomitant vaccine antigen.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population
Number analyzed (Participants) | 567 | 562
Percentage of participants
  Diphtheria toxoid: number analyzed (Participants) | 170 | 179
  Diphtheria toxoid | 85.0 [79.3 to 89.6] | 89.5 [84.4 to 93.4]
  Tetanus toxoid: number analyzed (Participants) | 191 | 197
  Tetanus toxoid | 95.5 [91.6 to 97.9] | 98.5 [95.7 to 99.7]
  Pertussis: PT: number analyzed (Participants) | 189 | 190
  Pertussis: PT | 94.5 [90.4 to 97.2] | 95.0 [91.0 to 97.6]
  Pertussis: FHA: number analyzed (Participants) | 187 | 190
  Pertussis: FHA | 93.5 [89.1 to 96.5] | 95.0 [91.0 to 97.6]
  Pertussis: PRN: number analyzed (Participants) | 187 | 190
  Pertussis: PRN | 93.5 [89.1 to 96.5] | 95.0 [91.0 to 97.6]
  Poliovirus: Type 1: number analyzed (Participants) | 91 | 102
  Poliovirus: Type 1 | 94.8 [88.3 to 98.3] | 98.1 [93.2 to 99.8]
  Poliovirus: Type 2: number analyzed (Participants) | 85 | 95
  Poliovirus: Type 2 | 88.5 [80.4 to 94.1] | 91.3 [84.2 to 96.0]
  Poliovirus: Type 3: number analyzed (Participants) | 92 | 104
  Poliovirus: Type 3 | 95.8 [89.7 to 98.9] | 100.0 [96.5 to 100.0]
  Hemophilus influenzae type b: number analyzed (Participants) | 207 | 193
  Hemophilus influenzae type b | 100.0 [98.2 to 100.0] | 100.0 [98.1 to 100.0]
Statistical Analysis 1: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Diphtheria; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = -4.5, 95% CI 2-sided [-11.2 to 2.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Tetanus; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = -3.0, 95% CI 2-sided [-7.0 to 0.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; PT; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = -0.5, 95% CI 2-sided [-5.2 to 4.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; FHA; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = -1.5, 95% CI 2-sided [-6.4 to 3.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; PRN; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = -1.5, 95% CI 2-sided [-6.4 to 3.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Poliovirus Type 1; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = -3.3, 95% CI 2-sided [-10.0 to 2.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Poliovirus Type 2; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = -2.8, 95% CI 2-sided [-11.8 to 5.8] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Poliovirus Type 3; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = -4.2, 95% CI 2-sided [-10.2 to -0.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: 20vPnC: Primary Study Population vs 13vPnC: Primary Study Population; Hib; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percent difference = 0.0, 95% CI 2-sided [-1.8 to 2.0] — [estimate comment as in outcome 14, analysis 1]

37. Secondary Outcome: Percentage of Participants With Predefined Pneumococcal IgG Antibody 1 Month After Dose 3: Russian Cohort
Description: as for outcome 32
Time Frame: 1 Month after Dose 3
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 22 | 24
Percentage of participants
  Serotype 1 | 90.9 [70.8 to 98.9] | 83.3 [62.6 to 95.3]
  Serotype 3 | 68.2 [45.1 to 86.1] | 50.0 [29.1 to 70.9]
  Serotype 4 | 95.5 [77.2 to 99.9] | 100.0 [85.8 to 100.0]
  Serotype 5 | 90.9 [70.8 to 98.9] | 91.7 [73.0 to 99.0]
  Serotype 6A | 95.5 [77.2 to 99.9] | 100.0 [85.8 to 100.0]
  Serotype 6B | 90.9 [70.8 to 98.9] | 91.7 [73.0 to 99.0]
  Serotype 7F | 95.5 [77.2 to 99.9] | 100.0 [85.8 to 100.0]
  Serotype 9V | 100.0 [84.6 to 100.0] | 83.3 [62.6 to 95.3]
  Serotype 14 | 90.9 [70.8 to 98.9] | 100.0 [85.8 to 100.0]
  Serotype 18C | 90.9 [70.8 to 98.9] | 95.8 [78.9 to 99.9]
  Serotype 19A | 100.0 [84.6 to 100.0] | 95.8 [78.9 to 99.9]
  Serotype 19F | 100.0 [84.6 to 100.0] | 91.7 [73.0 to 99.0]
  Serotype 23F | 90.9 [70.8 to 98.9] | 79.2 [57.8 to 92.9]
  Serotype 8 | 68.2 [45.1 to 86.1] | 25.0 [9.8 to 46.7]
  Serotype 10A | 68.2 [45.1 to 86.1] | 16.7 [4.7 to 37.4]
  Serotype 11A | 77.3 [54.6 to 92.2] | 20.8 [7.1 to 42.2]
  Serotype 12F | 36.4 [17.2 to 59.3] | 4.2 [0.1 to 21.1]
  Serotype 15B | 90.9 [70.8 to 98.9] | 20.8 [7.1 to 42.2]
  Serotype 22F | 63.6 [40.7 to 82.8] | 12.5 [2.7 to 32.4]
  Serotype 33F | 72.7 [49.8 to 89.3] | 20.8 [7.1 to 42.2]

38. Secondary Outcome: GMTs of Serotype-specific OPA at 1 Month After Dose 2: Russian Cohort
Description: as for outcome 33
Time Frame: 1 month after Dose 2
Population: Dose 2 evaluable immunogenicity population: eligible participants 42-70 days of age at first vaccination, received first 2 doses as randomized, at least 1 valid immunogenicity results from blood collection (27 to 56 days after Dose 2), no other major protocol deviations. "Number of participants Analyzed"= participants in Dose 2 evaluable immunogenicity population, ""Number Analyzed"= participants with valid OPA assay results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 24 | 27
Titers
  Serotype 1: number analyzed (Participants) | 8 | 9
  Serotype 1 | 17 [7 to 40] | 33 [10 to 105]
  Serotype 3: number analyzed (Participants) | 8 | 9
  Serotype 3 | 79 [42 to 149] | 31 [13 to 73]
  Serotype 4: number analyzed (Participants) | 8 | 9
  Serotype 4 | 166 [38 to 736] | 163 [32 to 840]
  Serotype 5: number analyzed (Participants) | 8 | 9
  Serotype 5 | 28 [11 to 76] | 31 [14 to 71]
  Serotype 6A: number analyzed (Participants) | 8 | 9
  Serotype 6A | 222 [32 to 1553] | 247 [60 to 1011]
  Serotype 6B: number analyzed (Participants) | 7 | 8
  Serotype 6B | 314 [27 to 3584] | 216 [39 to 1186]
  Serotype 7F: number analyzed (Participants) | 8 | 9
  Serotype 7F | 809 [481 to 1361] | 717 [246 to 2084]
  Serotype 9V: number analyzed (Participants) | 8 | 9
  Serotype 9V | 218 [70 to 676] | 293 [85 to 1008]
  Serotype 14: number analyzed (Participants) | 7 | 9
  Serotype 14 | 984 [492 to 1970] | 247 [69 to 886]
  Serotype 18C: number analyzed (Participants) | 8 | 9
  Serotype 18C | 968 [403 to 2326] | 268 [43 to 1655]
  Serotype 19A: number analyzed (Participants) | 7 | 9
  Serotype 19A | 314 [68 to 1443] | 31 [8 to 118]
  Serotype 19F: number analyzed (Participants) | 8 | 9
  Serotype 19F | 120 [27 to 529] | 230 [48 to 1097]
  Serotype 23F: number analyzed (Participants) | 8 | 9
  Serotype 23F | 35 [6 to 196] | 56 [9 to 346]
  Serotype 8: number analyzed (Participants) | 7 | 9
  Serotype 8 | 203 [19 to 2155] | 38 [9 to 161]
  Serotype 10A: number analyzed (Participants) | 6 | 5
  Serotype 10A | 559 [50 to 6233] | 232 [8 to 6478]
  Serotype 11A: number analyzed (Participants) | 6 | 7
  Serotype 11A | 3537 [863 to 14497] | 2717 [470 to 15716]
  Serotype 12F: number analyzed (Participants) | 7 | 9
  Serotype 12F | 698 [77 to 6301] | 198 [41 to 960]
  Serotype 15B: number analyzed (Participants) | 7 | 8
  Serotype 15B | 142 [9 to 2269] | 242 [18 to 3267]
  Serotype 22F: number analyzed (Participants) | 7 | 8
  Serotype 22F | 413 [32 to 5406] | 499 [28 to 8837]
  Serotype 33F: number analyzed (Participants) | 7 | 9
  Serotype 33F | 3508 [349 to 35250] | 3961 [706 to 22238]

39. Secondary Outcome: GMTs of Serotype-specific OPA at 1 Month After Dose 3: Russian Cohort
Description: as for outcome 34
Time Frame: 1 Month after Dose 3
Population: Dose 3 evaluable immunogenicity population = eligible participants 42-70 days of age at first vaccination, received all 3 doses as randomized with 335-455 days of age at Dose 3, at least 1 valid immunogenicity results from blood collection within 27 to 56 days after Dose 3, no major protocol deviations. "Number of participants Analyzed"= participants in Dose 3 evaluable immunogenicity population; "Number Analyzed"= participants with valid OPA assay results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
Number analyzed (Participants) | 22 | 24
Titers
  Serotype 1: number analyzed (Participants) | 8 | 9
  Serotype 1 | 85 [17 to 421] | 93 [22 to 394]
  Serotype 3: number analyzed (Participants) | 8 | 9
  Serotype 3 | 126 [41 to 383] | 107 [37 to 309]
  Serotype 4: number analyzed (Participants) | 8 | 8
  Serotype 4 | 310 [86 to 1123] | 429 [38 to 4863]
  Serotype 5: number analyzed (Participants) | 8 | 9
  Serotype 5 | 116 [28 to 476] | 108 [26 to 456]
  Serotype 6A: number analyzed (Participants) | 7 | 9
  Serotype 6A | 2922 [311 to 27459] | 1580 [393 to 6351]
  Serotype 6B: number analyzed (Participants) | 7 | 7
  Serotype 6B | 4417 [998 to 19951] | 1397 [150 to 12967]
  Serotype 7F: number analyzed (Participants) | 8 | 8
  Serotype 7F | 1039 [509 to 2122] | 1411 [373 to 5340]
  Serotype 9V: number analyzed (Participants) | 8 | 7
  Serotype 9V | 1574 [369 to 6711] | 1067 [150 to 7583]
  Serotype 14: number analyzed (Participants) | 7 | 9
  Serotype 14 | 1151 [321 to 4132] | 628 [137 to 2890]
  Serotype 18C: number analyzed (Participants) | 8 | 8
  Serotype 18C | 583 [149 to 2284] | 973 [89 to 10606]
  Serotype 19A: number analyzed (Participants) | 8 | 7
  Serotype 19A | 652 [131 to 3234] | 435 [14 to 13833]
  Serotype 19F: number analyzed (Participants) | 7 | 9
  Serotype 19F | 1570 [239 to 10337] | 701 [124 to 3958]
  Serotype 23F: number analyzed (Participants) | 8 | 8
  Serotype 23F | 152 [24 to 966] | 410 [22 to 7594]
  Serotype 8: number analyzed (Participants) | 4 | 6
  Serotype 8 | 368 [11 to 12078] | 149 [9 to 2337]
  Serotype 10A: number analyzed (Participants) | 4 | 6
  Serotype 10A | 2851 [1309 to 6210] | 117 [15 to 916]
  Serotype 11A: number analyzed (Participants) | 4 | 4
  Serotype 11A | 7137 [1036 to 49164] | 1789 [36 to 89068]
  Serotype 12F: number analyzed (Participants) | 4 | 7
  Serotype 12F | 757 [15 to 37522] | 241 [16 to 3734]
  Serotype 15B: number analyzed (Participants) | 5 | 7
  Serotype 15B | 822 [42 to 16070] | 147 [10 to 2214]
  Serotype 22F: number analyzed (Participants) | 4 | 7
  Serotype 22F | 1983 [390 to 10085] | 1635 [165 to 16157]
  Serotype 33F: number analyzed (Participants) | 3 | 7
  Serotype 33F | 5903 [53 to 657862] | 3619 [948 to 13817]

ADVERSE EVENTS:
Time Frame: Local reactions and Systemic events (systematic assessment): Within 7 days after Dose 1, 2, or 3; SAEs (non-systematic assessment): From Dose 1 up to 1 month after Dose 3 and other AEs (non-systematic assessment): From Dose 1 up to 1 month after Dose 2 and from Dose 3 up to 1 month after Dose 3
Description: Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. Event may be classified as serious in 1 participant and non-serious in another, or 1 participant may have experienced both during study. Safety analysis set evaluated. MedDRA 25.0 was used for primary cohorts and 26.0 was used for Russian cohort.
Arm/Group | 20vPnC: Primary Study Population | 13vPnC: Primary Study Population | 20vPnC: Russian Cohort | 13vPnC: Russian Cohort
All-Cause Mortality (participants affected / at risk) | 0/601 | 0/603 | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 34/601 | 40/603 | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 589/601 | 593/603 | 17/24 | 20/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20vPnC: Primary Study Population (N=601) | 13vPnC: Primary Study Population (N=603) | 20vPnC: Russian Cohort (N=24) | 13vPnC: Russian Cohort (N=27)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Thymus enlargement (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Aorticopulmonary septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Bronchogenic cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Bronchiolitis (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Bronchitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Erythema infectiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Gastroenteritis (Infections and infestations) | 4 (4) | 5 (5) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Gastrointestinal infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Herpangina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Laryngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Meningitis enteroviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (5) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Viral infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Underweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20vPnC: Primary Study Population (N=601) | 13vPnC: Primary Study Population (N=603) | 20vPnC: Russian Cohort (N=24) | 13vPnC: Russian Cohort (N=27)
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 345 (522) | 323 (465) | 9 (10) | 8 (10) — MedDRA 26.0 was used for Russian Cohorts.
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 495 (965) | 512 (970) | 8 (11) | 11 (16) — MedDRA 26.0 was used for Russian Cohorts.
Irritability (IRRITABILITY) (Psychiatric disorders) | 553 (1266) | 556 (1258) | 13 (18) | 15 (24) — MedDRA 26.0 was used for Russian Cohorts.
Injection site erythema (REDNESS) (General disorders) | 331 (534) | 333 (531) | 3 (4) | 4 (6) — MedDRA 26.0 was used for Russian Cohorts.
Injection site pain (PAIN) (General disorders) | 343 (555) | 347 (557) | 7 (8) | 6 (7) — MedDRA 26.0 was used for Russian Cohorts.
Injection site swelling (SWELLING) (General disorders) | 260 (431) | 251 (388) | 4 (5) | 3 (3) — MedDRA 26.0 was used for Russian Cohorts.
Pyrexia (FEVER) (General disorders) | 212 (282) | 214 (273) | 2 (3) | 4 (4) — MedDRA 26.0 was used for Russian Cohorts.
Upper respiratory tract infection (Infections and infestations) | 21 (21) | 35 (40) | 1 (1) | 0 (0) — MedDRA 26.0 was used for Russian Cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT04546425/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT04546425/SAP_001.pdf